CLINICAL TRIAL: NCT05131477
Title: A Phase IIb, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter Dose Ranging Study of a Subcutaneous Anti-OX40L Monoclonal Antibody (KY1005) in Moderate-to-Severe Atopic Dermatitis
Brief Title: Study Testing Response Effect of KY1005 Against Moderate-to-Severe Atopic Dermatitis, The STREAM-AD Study
Acronym: STREAM-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kymab Limited (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY1005-CT05/DRI17366; 2021-000725-28 (EudraCT Number); U1111-1271-1438 (Other: Universal Trial Number); DRI17366 (Other: Sponsor)
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Eczema; Atopic Dermatitis
Keywords: KY1005; Monoclonal Antibody; Atopic Dermatitis; Atopic Eczema; OX40L
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 250mg (500mg Loading Dose) KY1005 (Experimental): Every 4 weeks
  Interventions: Drug: Amlitelimab
- 250mg (No Loading Dose) KY1005 (Experimental): Every 4 weeks
  Interventions: Drug: Amlitelimab
- 125mg KY1005 (Experimental): Every 4 weeks
  Interventions: Drug: Amlitelimab
- 62.5mg KY1005 (Experimental): Every 4 weeks
  Interventions: Drug: Amlitelimab
- Placebo (Placebo Comparator): Every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Other Names: KY1005; SAR445229; A human anti-OX40 ligand monoclonal antibody
  Arms: 125mg KY1005; 250mg (500mg Loading Dose) KY1005; 250mg (No Loading Dose) KY1005; 62.5mg KY1005
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
This is an interventional, randomized, parallel group, treatment, Phase IIb, double blind, 5-arm study to assess the effect of Anti-OX40L Monoclonal Antibody (KY1005) in adult participants with moderate to severe atopic dermatitis.

The estimated duration is 28 days for screening and then up to approximately day 477 (last dose no later than day 337+140 days safety follow-up) for all patients unless enrolled into the Long-Term Extension (LTE) protocol (NCT05492578) at either Day 169 depending on responder status or no later than Day 365 due to loss of clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to < 75 years of age) with AD as defined by the American Academy of Dermatology Consensus Criteria for 1 year or longer at Baseline.
* Eczema Area and Severity Index (EASI) of 12 or higher at the Screening Visit and 16 or higher at Baseline.
* Investigator's Global Assessment (IGA) Scale of 3 or 4 at Baseline.
* AD involvement of 10% or more of body surface area (BSA) at Baseline.
* Baseline worst/maximum pruritus Numeric Rating Scale (NRS) of ≥4.
* Documented history, within 6 months prior to Baseline, of either inadequate response or inadvisability of topical treatments.
* Must have applied a stable dose of topical bland emollient (simple moisturizer, no additives [e.g., urea]) at least twice daily for a minimum of 7 consecutive days before Baseline.
* Able to complete patient questionnaires.
* Able and willing to comply with requested study visits/telephone visits and procedures.
* Able and willing to provide written informed consent.
* For patients who decide to join the biopsy sub-study be able and willing to provide skin biopsies.

Exclusion Criteria:

* Treatment within specific time windows before the baseline visit for the management of atopic dermatitis such as topical or systemic corticosteroids, biologic or investigational therapies and/or phototherapy.
* Known history of, or suspected, significant current immunosuppression, including history of invasive opportunistic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Weight <40 kg or >150 kg at Baseline.
* Treatment with a live (attenuated) immunization within 12 weeks prior to Baseline.
* Men and women (of reproductive potential) unwilling to use birth control and women who are pregnant or breastfeeding.
* Any malignancies or history of malignancies prior to Baseline (except for non-melanoma skin cancer that has been excised and cured for more than 3 years prior to Baseline; in situ cervical carcinoma that has been excised and cured).
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C at the screening visit.
* Severe concomitant illness that would in the Investigator's opinion inhibit the patient's participation in the study, including for example, but not limited to, hypertension, renal disease, neurological conditions, heart failure and pulmonary disease.
* In the Investigator's opinion, any clinically significant laboratory results from the clinical chemistry, hematology or urinalysis tests at the Screening Visit.
* Concurrent participation in any other clinical study, including non-interventional studies.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (20):
  - Investigative Site Number: 1018, Fremont, California
  - Investigative site #1022, Sacramento, California
  - Investigative Site Number: 1006, Boca Raton, Florida
  - Investigative Site Number: 1001, Clearwater, Florida
  - Investigative Site Number: 1019, Coral Gables, Florida
  - Investigative Site Number: 1007, Miami, Florida
  - Investigative Site Number: 1013, Tampa, Florida
  - Investigative Site Number: 1004, Savannah, Georgia
  - Investigative Site Number: 1010, Clarksville, Indiana
  - Investigative Site Number: 1015, Indianapolis, Indiana
  - Investigative Site Number: 1021, Louisville, Kentucky
  - Investigative Site Number: 1011, Towson, Maryland
  - Investigative Site Number: 1014, Beverly, Massachusetts
  - Investigative Site Number: 1012, Troy, Michigan
  - Investigative Site Number: 1005, Tulsa, Oklahoma
  - Investigative Site Number: 1017, Portland, Oregon
  - Investigative Site Number: 1009, Portland, Oregon
  - Investigative Site Number: 1003, Anderson, South Carolina
  - Investigative Site Number: 1008, Murfreesboro, Tennessee
  - Investigative site #1023, Mansfield, Texas
- Australia (3):
  - Investigative Site Number 3002, Carlton
  - Investigative Site Number: 3003, East Melbourne
  - Investigational Site Number: 3001, Parkville
- Bulgaria (6):
  - Investigative Site Number: 2004, Pleven
  - Investigative Site Number: 2005, Sofia
  - Investigative Site Number: 2006, Sofia
  - Investigative Site Number: 2003, Sofia
  - Investigative Site Number: 2002, Sofia
  - Investigative Site Number: 2001, Stara Zagora
- Canada (5):
  - Investigative Site Number: 1106, Markham, Ontario
  - Investigative site #1108, Niagara Falls, Ontario
  - Investigative Site Number: 1103, Ottawa, Ontario
  - Investigative Site Number: 1107, Waterloo, Ontario
  - Investigative Site Number: 1101, Windsor, Ontario
- Czechia (6):
  - Investigative Site Number: 2105, Nový Jicín, Moravskoslezský kraj
  - Investigative Site Number: 2102, Prague, Praha, Hlavní Mesto
  - Investigative Site Number: 2103, Prague, Praha, Hlavní Mesto
  - Investigative Site Number: 2108, Brno, South Moravian
  - Investigative Site Number: 2106, Kutná Hora
  - Investigative Site Number: 2104, Ostrava
- Germany (6):
  - Investigative Site Number: 2209, Erlangen, Bavaria
  - Investigative Site Number: 2202, Blankenfelde, Brandenburg
  - Investigator Site Number: 2201, Münster, North Rhine-Westphalia
  - Investigative Site Number: 2208, Kiel, Schleswig-Holstein
  - Investigative Site Number: 2203, Berlin
  - Investigative Site Number: 2204, Hamburg
- Hungary (7):
  - Investigative Site Number: 2305, Gyula, Bekes County
  - Investigative Site Number: 2307, Kecskemét, Bács-Kiskun county
  - Investigative Site Number: 2301, Szeged, Csongrád megye
  - Investigative Site Number: 2303, Debrecen, Hajdú-Bihar
  - Investigative Site Number: 2306, Szolnok, Jász-Nagykun-Szolnok
  - Investigative Site Number: 2302, Zalaegerszeg, Zala County
  - Investigative Site Number: 2304, Budapest
- Japan (15):
  - Investigative Site Number: 3103, Matsudo, Chiba
  - Investigative Site Number: 3114, Obihiro-Shi, Hokkaidô
  - Investigative site #3108, Kagoshima, Kagoshima-ken
  - Investigative site #3113, Yokohama, Kanagawa
  - Investigative Site Number: 3112, Adachi-Ku, Tokyo
  - Investigative Site Number: 3115, Chuo Ku, Tokyo
  - Investigative Site Number: 3104, Edagowa-Ku, Tokyo
  - Investigative Site Number: 3111, Koto-Ku, Tokyo
  - Investigative Site Number: 3107, Minato-Ku, Tokyo
  - Investigative site #3105, Setagaya-Ku, Tokyo
  - Investigative site #3102, Kyoto
  - Investigative Site Number: 3106, Mibu-machi
  - Investigative site #3101, Sapporo
  - Investigative Site Number: 3109, Habikino-Shi, Ôsaka
  - Investigative Site Number: 3110, Sakaishi, Ôsaka
- Poland (22):
  - Investigative Site Number: 2408, Krakow, Lesser Poland Voivodeship
  - Investigative Site Number: 2407, Krakow, Lesser Poland Voivodeship
  - Investigative Site Number: 2409, Krakow, Lesser Poland Voivodeship
  - Investigative Site Number: 2414, Wroclaw, Lower Silesian Voivodeship
  - Investigative Site Number: 2418, Wroclaw, Lower Silesian Voivodeship
  - Investigative Site Number: 2417, Wroclaw, Lower Silesian Voivodeship
  - Investigative Site Number: 2420, Lodz, Lódzkie
  - Investigative Site Number: 2415, Lódz, Lódzkie
  - Investigative Site Number: 2412, Warsaw, Masovian Voivodeship
  - Investigative Site Number: 2411, Warsaw, Masovian Voivodeship
  - Investigative Site Number: 2413, Warsaw, Masovian Voivodeship
  - Investigative Site Number: 2401, Rzeszów, Podkarpackie Voivodeship
  - Investigative site #2419, Bialystok, Podlaskie Voivodeship
  - Investigative Site Number: 2402, Gdansk, Pomeranian Voivodeship
  - Investigative Site Number: 2404, Gdynia, Pomeranian Voivodeship
  - Investigative Site Number: 2405, Katowice, Silesian Voivodeship
  - Investigative Site Number: 2410, Szczecin, West Pomeranian Voivodeship
  - Investigative site #2419, Bialystok
  - Investigative Site Number: 2403, Gdansk
  - Investigative Site Number: 2406, Krakow
  - Investigative site #2420, Lodz
  - Investigative Site Number: 2416, Lodz, Łódź Voivodeship
- Spain (5):
  - Investigative Site Number: 2502, Manises, Valencia
  - Investigative Site Number: 2505, Alicante
  - Investigative Site Number: 2501, Córdoba
  - Investigative Site Number: 2503, Madrid
  - Investigative Site Number: 2504, Pontevedra
- Taiwan (4):
  - Investigative Site Number: 3201, Niao Song Qu
  - Investigative Site Number: 3202, Taichung
  - Investigative site # 3206, Taipei
  - Investigative Site Number: 3203, Taoyuan District
- United Kingdom (3):
  - Investigative Site Number: 2603, London
  - Investigative Site Number: 2601, London
  - Investigative Site Number: 2602, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.
  Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org
Supporting Information: Study Protocol, SAP
URL: https://vivli.org

REFERENCES:
- [Derived] Reich A, Blauvelt A, Weidinger S, Shi VY, Katoh N, Lynde C, Gao X, Armstrong NM, Bernigaud C, Rahawi K. A Post Hoc Analysis of Atopic Dermatitis of the Head and Neck and Other Body Regions from the Amlitelimab STREAM-AD Phase 2b Study. Dermatol Ther (Heidelb). 2025 Dec 8. doi: 10.1007/s13555-025-01609-6. Online ahead of print. PMID 41359216
- [Derived] Blauvelt A, Chovatiya R, Merola JF, Weidinger S, Igawa K, Brookes E, Weber C, Wang J, Gray C. Improvement and maintenance of clinical outcome assessments in atopic dermatitis with amlitelimab. J Eur Acad Dermatol Venereol. 2025 Dec;39(12):2113-2120. doi: 10.1111/jdv.20877. Epub 2025 Jul 24. PMID 40704660
- [Derived] Weidinger S, Blauvelt A, Papp KA, Reich A, Lee CH, Worm M, Lynde C, Kataoka Y, Foley P, Wei X, Wong W, Solente AC, Weber C, Adelman S, Davey S, Hurbin F, Rynkiewicz N, Yen K, O'Malley JT, Bernigaud C. Phase 2b randomized clinical trial of amlitelimab, an anti-OX40 ligand antibody, in patients with moderate-to-severe atopic dermatitis. J Allergy Clin Immunol. 2025 Apr;155(4):1264-1275. doi: 10.1016/j.jaci.2024.10.031. Epub 2024 Nov 8. PMID 39522654
- See also: DRI17366 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25401&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started in December 2021 and ended in February 2024. An individual participant was part of this study for about 1 year and 5 months. The study took place at 100 sites in 12 countries. Up to 350 participants (approximately 70 participants per treatment group) were planned to be enrolled.
Pre-assignment Details: The study was performed in 2 parts: Part 1 for all population (baseline to Week 24) for efficacy and safety and Part 2 for Part 1 Responders (Week 24 to Week 52 for efficacy and Week 24 to Week 68 for safety). Responders are defined as participants who achieved ≥EASI 75 and/or IGA 0/1 at Week 24.
Groups:
- 250 mg (500 mg LD) KY1005 (Part 1): Participants randomized to receive 500 mg loading dose of KY1005 at baseline, followed 4 weeks later with 250 mg of KY1005 every 4 weeks (Q4W) injection for 24 weeks.
- 250 mg (no LD) KY1005 (Part 1): Participants randomized to receive 250 mg (as injection) plus placebo at baseline, followed 4 weeks later with 250 mg Q4W as injection for 24 weeks.
- 125 mg KY1005 (Part 1): Participants randomized to receive 125 mg (as injection) plus placebo at baseline, followed 4 weeks later with 125 mg Q4W as injection for 24 weeks.
- 62.5 mg KY1005 (Part 1): Participants randomized to receive 62.5 mg (as injection) plus placebo at baseline, followed 4 weeks later with 62.5 mg Q4W as injection for 24 weeks.
- Placebo (Part 1): Participants randomized to receive placebo given as injections at baseline, followed 4 weeks later with placebo (0 mg) Q4W as injection for 24 weeks.
- 250 mg KY1005 Re-Randomized From the 250 mg (LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (500 mg LD) at Part 1) were re-randomized to receive KY1005 250mg Q4W from Week 24 to Week 52
- Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (500 mg LD) at Part 1) were re-randomized to receive placebo Q4W from Week 24 to Week 52
- 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (no LD) at Part 1) were rerandomized to receive KY1005 250mg Q4W from Week 24 to Week 52
- Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (no LD) at Part 1) were rerandomized to receive placebo Q4W from Week 24 to Week 52
- 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 125 mg at Part 1) were rerandomized to receive KY1005 125 mg Q4W from Week 24 to Week 52
- Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 125 mg at Part 1) were rerandomized to receive placebo Q4W from Week 24 to Week 52
- 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (62.5 mg) were re-randomized to receive KY1005 62.5mg Q4W from Week 24 to Week 52
- Placebo Re-randomized From the 62.5 mg Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 62.5 mg at Part 1) were rerandomized to receive placebo Q4W from Week 24 to Week 52
- Placebo (Part 2) Continued From Part 1 Placebo: Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) placebo received placebo Q4W from Week 24 to Week 52
Period: PART 1
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1) | 250 mg KY1005 Re-Randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Started (Randomized) | 77 | 78 | 77 | 79 | 79 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Randomized and Treated | 77 | 78 | 77 | 78 | 78 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Re-randomized at Week 24 | 47 | 40 | 45 | 42 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 68 | 62 | 69 | 67 | 57 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 16 | 8 | 12 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 9 | 6 | 2 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 5 | 1 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — unclassified | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized and not treated | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PART 2
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1) | 250 mg KY1005 Re-Randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Started | 0 | 0 | 0 | 0 | 0 | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Re-randomized and Treated | 0 | 0 | 0 | 0 | 0 | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 34 | 15
Completed | 0 | 0 | 0 | 0 | 0 | 12 | 31 | 11 | 24 | 11 | 28 | 7 | 29 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 4 | 1 | 5 | 0 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 2 | 0
Not completed — Unclassified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Re-randomized and not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (No LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1) | Total
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (13.32) | 40.8 (15.24) | 37.9 (15.17) | 37.6 (14.78) | 36.4 (13.07) | 37.8 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 39 | 37 | 30 | 171
  Male | 47 | 43 | 38 | 42 | 49 | 219
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were 390 participants enrolled in Part 1 and 190 participants enrolled in Part 2.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 12 | 12 | 10 | 14 | 12 | 60
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 4 | 2 | 4 | 4 | 6 | 20
    White | 61 | 63 | 63 | 60 | 60 | 307
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 3
EASI Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — Eczema Area and Severity Index-The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD with scores from 0 to 72. Higher scores indicate worse condition.
  units on a scale | 30.3 (11.66) | 28.7 (10.53) | 30.3 (12.43) | 28.7 (10.09) | 26.4 (7.85) | 28.9 (10.65)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in EASI (Eczema Area and Severity Index) From Baseline to Week 16 (Part 1)
Description: Eczema Area and Severity Index-The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD with scores from 0 to 72. Higher scores indicate worse condition.
Time Frame: Baseline to week 16
Population: Full Analysis Set for Part 1. The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. Efficacy analyses were based on treatment allocated at randomization. The Primary efficacy endpoint is the percentage of change in EASI from Baseline to Day 113 (Week 16). The primary analysis was conducted on FAS1 after all the randomized patients had reached the Day 169 (Week 24) visit/ early termination. Missing data were imputed by multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
percentage of change | -61.5 (4.68) | -56.8 (4.59) | -51.6 (4.59) | -59.6 (4.53) | -29.4 (4.76)
Statistical Analysis 1: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -32.1, 95% CI 2-sided [-43.9 to -20.3], Standard Error of Mean 6.01 — LS Mean Difference
Statistical Analysis 2: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -27.3, 95% CI 2-sided [-39.1 to -15.6], Standard Error of Mean 5.98 — LS Mean Difference
Statistical Analysis 3: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -22.2, 95% CI 2-sided [-34.0 to -10.4], Standard Error of Mean 6.01 — LS Mean Difference
Statistical Analysis 4: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -30.2, 95% CI 2-sided [-41.9 to -18.5], Standard Error of Mean 5.95

2. Secondary Outcome: Percentage Change in EASI (Eczema Area and Severity Index) From Baseline to Week 24 (Part 1)
Description: as for outcome 1
Time Frame: Baseline to week 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. The primary analysis was conducted on the FAS1 after all randomized patients had reached day 169 (Week 24) visit/ early termination. Percentage change from baseline in EASI at Day 169 (Week 24). Missing data were imputed by multiple imputation.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
percentage of change | -64.4 (5.17) | -52.2 (5.14) | -53.7 (5.08) | -54.4 (5.09) | -27.6 (5.29)
Statistical Analysis 1: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -36.8, 95% CI 2-sided [-49.8 to -23.8], Standard Error of Mean 6.62 — LS Mean Difference
Statistical Analysis 2: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -24.6, 95% CI 2-sided [-37.7 to -11.6], Standard Error of Mean 6.67 — LS Mean Difference
Statistical Analysis 3: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -26.2, 95% CI 2-sided [-39.2 to -13.1], Standard Error of Mean 6.65 — LS Mean Difference
Statistical Analysis 4: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -26.8, 95% CI 2-sided [-39.7 to -13.9], Standard Error of Mean 6.58 — LS Mean Difference

3. Secondary Outcome: Percentage of Participants With at Least a 75% Reduction From Baseline in EASI (EASI 75) at Week 16 and Week 24 (Part 1)
Description: as for outcome 1
Time Frame: Baseline to week 16 and week 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. The primary analysis was conducted on the FAS1 after all randomized patients had reached day 169 (Week 24) visit/ early termination. Percentage of patients with at least 75% reduction from baseline in EASI (EASI 5) at days 113 (Week 16) and Day 169 (Week 24). Participants with missing data were considered as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 16 | 40.3 | 38.5 | 42.9 | 40.5 | 11.4
  Week 24 | 54.5 | 38.5 | 49.4 | 40.5 | 17.7
Statistical Analysis 1: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.29, 95% CI 2-sided [0.16 to 0.42]
Statistical Analysis 2: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.27, 95% CI 2-sided [0.14 to 0.40]
Statistical Analysis 3: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.31, 95% CI 2-sided [0.18 to 0.44]
Statistical Analysis 4: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.29, 95% CI 2-sided [0.16 to 0.42]
Statistical Analysis 5: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.36, 95% CI 2-sided [0.23 to 0.5]
Statistical Analysis 6: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p = 0.0040, Cochran-Mantel-Haenszel; Proportion Difference = 0.21, 95% CI 2-sided [0.07 to 0.34]
Statistical Analysis 7: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.31, 95% CI 2-sided [0.17 to 0.45]
Statistical Analysis 8: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Test type: Superiority; p = 0.0016, Cochran-Mantel-Haenszel; Proportion Difference = 0.23, 95% CI 2-sided [0.09 to 0.36]

4. Secondary Outcome: Percentage of Participants With a Response of IGA (Investigator Global Assessment) 0 or 1 and a Reduction From Baseline ≥ 2 Points (Part 1)
Description: The IGA is a five-point scale that provides a global clinical assessment of AD severity ranging from 0 to 4, where 0 indicates clear,1 is almost clear, 2 is mild, 3 is moderate, and 4 indicates severe AD.
Time Frame: Baseline to week 16 and week 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. The primary analysis was conducted on the FAS1 after all randomized patients had reached day 169 (Week 24) visit/ early termination. Percentage of patients with a response of IGA 0 or 1 and a reduction from baseline of ≥ 2 points at Days 113 (Week 16) and Day 169 (Week 24). Participants with missing data were considered as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 16 | 22.1 | 14.1 | 19.5 | 25.3 | 5.1
  Week 24 | 45.5 | 33.3 | 40.3 | 29.1 | 11.4
Statistical Analysis 1: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel; Proportion Difference = 0.17, 95% CI 2-sided [0.06 to 0.27]
Statistical Analysis 2: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0562, Cochran-Mantel-Haenszel; Proportion Difference = 0.09, 95% CI 2-sided [0 to 0.18]
Statistical Analysis 3: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0054, Cochran-Mantel-Haenszel; Proportion Difference = 0.14, 95% CI 2-sided [0.04 to 0.24]
Statistical Analysis 4: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Proportion Difference = 0.2, 95% CI 2-sided [0.1 to 0.31]
Statistical Analysis 5: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.34, 95% CI 2-sided [0.21 to 0.47]
Statistical Analysis 6: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel; Proportion Difference = 0.22, 95% CI 2-sided [0.1 to 0.34]
Statistical Analysis 7: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 0.29, 95% CI 2-sided [0.16 to 0.41]
Statistical Analysis 8: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel; Proportion Difference = 0.18, 95% CI 2-sided [0.06 to 0.3]

5. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Weekly Average of Pruritus NRS (Numerical Rating Scale) ≥ 4 With a Baseline Pruritus of ≥ 4 From Baseline (Part 1)
Description: The pruritus NRS is a simple assessment tool to report the intensity of their pruritus (itch) ranges from 0 to 10 with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Time Frame: Baseline to week 16 and week 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. The primary analysis was conducted on the FAS1 after all randomized patients had reached day 169 (Week 24) visit/ early termination. Proportion of patients with improvement (reduction) of weekly average of pruritus NRS ≥ 4 a baseline pruritus NRS of ≥ 4 from baseline to Days 113 (Week 16) and Day 169 (Week 24). Participants with missing data were considered as non-responders.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo (Part 1): Participants randomized to receive 62.5 mg (as injection) plus placebo at baseline, followed 4 weeks later with 62.5 mg Q4W as injection for 24 weeks.
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 16 | 24.7 | 19.2 | 20.8 | 22.8 | 5.1
  Week 24 | 31.2 | 24.4 | 28.6 | 27.8 | 7.6
Statistical Analysis 1: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Proportion Difference = 0.19, 95% CI 2-sided [0.09 to 0.3]
Statistical Analysis 2: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0057, Cochran-Mantel-Haenszel; Proportion Difference = 0.14, 95% CI 2-sided [0.04 to 0.24]
Statistical Analysis 3: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0038, Cochran-Mantel-Haenszel; Proportion Difference = 0.16, 95% CI 2-sided [0.05 to 0.26]
Statistical Analysis 4: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Week 16; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel; Proportion Difference = 0.18, 95% CI 2-sided [0.07 to 0.28]
Statistical Analysis 5: Comparison: 250 mg (500 mg LD) KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Proportion Difference = 0.23, 95% CI 2-sided [0.11 to 0.35]
Statistical Analysis 6: Comparison: 250 mg (no LD) KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p = 0.0038, Cochran-Mantel-Haenszel; Proportion Difference = 0.17, 95% CI 2-sided [0.06 to 0.28]
Statistical Analysis 7: Comparison: 125 mg KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Proportion Difference = 0.21, 95% CI 2-sided [0.09 to 0.32]
Statistical Analysis 8: Comparison: 62.5 mg KY1005 (Part 1) vs Placebo (Part 1); Week 24; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel; Proportion Difference = 20, 95% CI 2-sided [9 to 32]

6. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Weekly Average of Pruritus NRS (Numerical Rating Scale) ≥ 4 With a Baseline Pruritus of ≥ 4 From Baseline (Part 2)
Description: as for outcome 5
Time Frame: Baseline to weeks week 24, 25, 26, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 38, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, 51, & 52
Population: The Full Analysis Set (FAS2) for Part 2 included all re-randomized at week 24. Only those participants with data available at specified time points are reported. Participants with missing data were considered as non-responders.
Measure: Number; unit: Percentage of participants
Groups:
- 250 mg KY1005 Re-Randomized From the LD Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (500 mg LD) at Part 1) were re-randomized to receive KY1005 250mg Q4W from Week 24 to Week 52
Arm/Group | 250 mg KY1005 Re-Randomized From the LD Arm (Part 2) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of participants
  Week 24 | 53.8 | 41.2 | 75.0 | 35.7 | 58.3 | 45.5 | 71.4 | 45.7 | 25.0
  Week 25 | 53.8 | 41.2 | 66.7 | 39.3 | 66.7 | 39.4 | 57.1 | 37.1 | 31.3
  Week 26 | 53.8 | 38.2 | 66.7 | 32.1 | 58.3 | 33.3 | 71.4 | 42.9 | 25.0
  Week 27 | 61.5 | 35.3 | 58.3 | 28.6 | 58.3 | 39.4 | 71.4 | 37.1 | 25.0
  Week 28 | 61.5 | 35.3 | 66.7 | 35.7 | 58.3 | 42.4 | 57.1 | 37.1 | 25.0
  Week 29 | 69.2 | 38.2 | 50.0 | 25.0 | 58.3 | 45.5 | 57.1 | 40.0 | 25.0
  Week 30 | 61.5 | 44.1 | 58.3 | 25.0 | 66.7 | 36.4 | 42.9 | 42.9 | 18.8
  Week 31 | 61.5 | 41.2 | 58.3 | 25.0 | 66.7 | 36.4 | 42.9 | 40.0 | 18.8
  Week 32 | 61.5 | 47.1 | 50.0 | 25.0 | 75.0 | 42.4 | 71.4 | 40.0 | 18.8
  Week 33 | 61.5 | 47.1 | 58.3 | 28.6 | 58.3 | 42.4 | 71.4 | 40.0 | 18.8
  Week 34 | 61.5 | 41.2 | 75.0 | 21.4 | 75.0 | 30.3 | 42.9 | 37.1 | 25.0
  Week 35 | 61.5 | 41.2 | 66.7 | 21.4 | 66.7 | 39.4 | 71.4 | 34.3 | 25.0
  Week 36 | 61.5 | 38.2 | 58.3 | 21.4 | 66.7 | 42.4 | 71.4 | 40.0 | 25.0
  Week 37 | 53.8 | 41.2 | 50.0 | 28.6 | 66.7 | 42.4 | 71.4 | 37.1 | 18.8
  Week 38 | 53.8 | 35.3 | 50.0 | 25.0 | 58.3 | 42.4 | 71.4 | 31.4 | 18.8
  Week 39 | 53.8 | 41.2 | 50.0 | 25.0 | 58.3 | 39.4 | 71.4 | 31.4 | 25.0
  Week 40 | 53.8 | 38.2 | 33.3 | 25.0 | 58.3 | 36.4 | 28.6 | 31.4 | 25.0
  Week 41 | 61.5 | 35.3 | 41.7 | 28.6 | 66.7 | 39.4 | 57.1 | 34.3 | 31.3
  Week 42 | 53.8 | 38.2 | 50.0 | 28.6 | 66.7 | 36.4 | 42.9 | 31.4 | 25.0
  Week 43 | 53.8 | 35.3 | 50.0 | 28.6 | 58.3 | 36.4 | 42.9 | 34.3 | 31.3
  Week 44 | 61.5 | 38.2 | 41.7 | 21.4 | 75.0 | 39.4 | 42.9 | 37.1 | 25.0
  Week 45 | 61.5 | 41.2 | 41.7 | 21.4 | 75.0 | 36.4 | 42.9 | 40.0 | 31.3
  Week 46 | 53.8 | 44.1 | 50.0 | 28.6 | 50.0 | 27.3 | 42.9 | 37.1 | 31.3
  Week 47 | 46.2 | 38.2 | 33.3 | 28.6 | 58.3 | 30.3 | 42.9 | 45.7 | 25.0
  Week 48 | 38.5 | 35.3 | 41.7 | 28.6 | 66.7 | 27.3 | 57.1 | 37.1 | 25.0
  Week 49 | 38.5 | 41.2 | 50.0 | 35.7 | 66.7 | 30.3 | 57.1 | 40.0 | 25.0
  Week 50 | 38.5 | 35.3 | 50.0 | 32.1 | 66.7 | 24.2 | 57.1 | 37.1 | 25.0
  Week 51 | 30.8 | 32.4 | 41.7 | 28.6 | 58.3 | 27.3 | 42.9 | 34.3 | 25.0
  Week 52 | 46.2 | 29.4 | 41.7 | 25.0 | 66.7 | 27.3 | 57.1 | 40.0 | 25.0

7. Secondary Outcome: Absolute Change From Baseline in EASI (Eczema Area and Severity Index) (Part 1)
Description: as for outcome 1
Time Frame: Baseline to weeks 2, 4, 8, 12, 16, 20 and 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. Only those participants with data available at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
score on a scale
  Week 2: number analyzed (Participants) | 73 | 77 | 75 | 75 | 78
  Week 2 | -8.49 (10.777) | -5.27 (8.485) | -6.17 (10.071) | -7.51 (8.836) | -3.98 (7.855)
  Week 4: number analyzed (Participants) | 76 | 74 | 76 | 77 | 75
  Week 4 | -11.21 (10.612) | -8.38 (9.944) | -10.33 (10.861) | -10.27 (10.550) | -7.20 (8.510)
  Week 8: number analyzed (Participants) | 70 | 70 | 75 | 76 | 72
  Week 8 | -15.67 (11.872) | -11.93 (11.018) | -13.77 (12.964) | -14.37 (10.054) | -7.64 (10.450)
  Week 12: number analyzed (Participants) | 70 | 70 | 72 | 77 | 70
  Week 12 | -18.49 (12.411) | -13.84 (11.121) | -16.56 (14.062) | -16.46 (11.699) | -8.76 (9.608)
  Week 16: number analyzed (Participants) | 70 | 69 | 73 | 76 | 69
  Week 16 | -19.71 (12.731) | -16.31 (12.329) | -15.70 (14.226) | -17.82 (11.730) | -7.47 (11.338)
  Week 20: number analyzed (Participants) | 67 | 69 | 72 | 72 | 67
  Week 20 | -21.93 (14.283) | -16.46 (12.834) | -16.98 (15.321) | -16.76 (12.590) | -7.91 (11.163)
  Week 24: number analyzed (Participants) | 71 | 68 | 72 | 70 | 67
  Week 24 | -21.92 (14.475) | -15.72 (12.977) | -16.91 (15.085) | -17.09 (13.088) | -7.52 (12.537)

8. Secondary Outcome: Percentage Change From Baseline in EASI (Eczema Area and Severity Index) (Part 1)
Description: as for outcome 1
Time Frame: Baseline to weeks 2,4, 8,12,16, 20 and 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. Only those participants with data available at specified time points are reported.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of change
  Week 2: number analyzed (Participants) | 73 | 77 | 75 | 75 | 78
  Week 2 | -27.94 (30.032) | -17.75 (38.988) | -19.09 (39.499) | -26.03 (34.462) | -15.26 (34.143)
  Week 4: number analyzed (Participants) | 76 | 74 | 76 | 77 | 75
  Week 4 | -36.85 (28.901) | -29.13 (42.013) | -35.10 (34.457) | -35.49 (38.786) | -27.56 (31.037)
  Week 8: number analyzed (Participants) | 70 | 70 | 75 | 76 | 72
  Week 8 | -50.25 (30.666) | -41.21 (41.129) | -45.96 (38.150) | -51.70 (31.046) | -28.70 (38.603)
  Week 12: number analyzed (Participants) | 70 | 70 | 72 | 77 | 70
  Week 12 | -59.61 (30.717) | -50.15 (36.086) | -55.23 (40.218) | -57.36 (34.275) | -33.72 (35.358)
  Week 16: number analyzed (Participants) | 70 | 69 | 73 | 76 | 69
  Week 16 | -62.35 (32.322) | -59.98 (37.444) | -52.50 (40.820) | -61.51 (31.663) | -28.25 (41.173)
  Week 20: number analyzed (Participants) | 67 | 69 | 72 | 72 | 67
  Week 20 | -67.85 (33.135) | -57.80 (38.921) | -56.29 (43.103) | -57.87 (38.977) | -30.32 (40.486)
  Week 24: number analyzed (Participants) | 71 | 68 | 72 | 70 | 67
  Week 24 | -68.01 (36.052) | -55.84 (40.299) | -56.72 (44.271) | -57.37 (40.225) | -28.55 (44.004)

9. Secondary Outcome: Absolute Change From Baseline in EASI (Eczema Area and Severity Index) (Part 2)
Description: as for outcome 1
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48, & 52
Population: The Full Analysis Set (FAS2) for Part 2 included all re-randomized at week 24. Only those participants with data available at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg KY1005 Re-Randomized From the LD Arm (Part 2) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Score on a scale
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 5 | 33 | 16
  Week 24 | -29.65 (11.278) | -26.28 (13.353) | -27.60 (11.170) | -18.90 (11.932) | -27.10 (12.670) | -22.45 (14.998) | -25.47 (12.209) | -22.41 (12.841) | -21.47 (10.420)
  Week 28: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 7 | 34 | 14
  Week 28 | -30.51 (12.422) | -26.34 (14.353) | -25.86 (13.128) | -17.29 (12.458) | -26.37 (13.067) | -22.87 (15.667) | -23.79 (10.424) | -21.75 (13.106) | -21.69 (11.918)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -29.08 (14.544) | -24.79 (15.775) | -22.99 (15.741) | -15.38 (12.620) | -27.36 (13.383) | -22.94 (14.915) | -24.94 (11.245) | -20.32 (14.189) | -19.60 (10.632)
  Week 36: number analyzed (Participants) | 13 | 33 | 10 | 28 | 12 | 32 | 7 | 32 | 15
  Week 36 | -28.15 (15.138) | -22.78 (17.505) | -22.27 (16.368) | -14.57 (13.550) | -27.51 (13.550) | -22.99 (14.978) | -24.65 (10.801) | -20.09 (15.098) | -20.20 (10.436)
  Week 40: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 32 | 7 | 31 | 15
  Week 40 | -28.54 (15.203) | -22.30 (17.908) | -22.56 (14.949) | -14.81 (13.178) | -27.96 (14.444) | -20.45 (16.659) | -25.51 (11.796) | -20.80 (14.601) | -20.05 (10.596)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -28.43 (15.061) | -22.23 (17.487) | -23.07 (15.679) | -14.49 (12.877) | -27.49 (14.324) | -19.76 (16.561) | -22.34 (11.070) | -20.70 (14.343) | -20.43 (11.007)
  Week 48: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -22.15 (14.876) | -21.82 (17.764) | -22.24 (16.312) | -13.95 (13.596) | -27.72 (14.882) | -18.34 (16.959) | -23.88 (12.517) | -19.74 (15.277) | -19.99 (11.292)
  Week 52: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 29 | 7 | 31 | 14
  Week 52 | -22.03 (14.889) | -19.59 (15.321) | -22.68 (15.418) | -13.89 (13.427) | -28.08 (16.097) | -17.30 (16.752) | -23.26 (11.789) | -20.81 (14.813) | -20.30 (11.526)

10. Secondary Outcome: Percentage Change From Baseline in EASI (Eczema Area and Severity Index) (Part 2)
Description: as for outcome 1
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48, & 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg KY1005 Re-Randomized From the LD Arm (Part 2) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of change
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 5 | 33 | 16
  Week 24 | -91.71 (8.539) | -81.85 (31.624) | -84.20 (16.741) | -72.72 (41.299) | -90.91 (10.585) | -74.56 (39.811) | -85.81 (10.212) | -76.74 (30.922) | -78.51 (28.977)
  Week 28: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 7 | 34 | 14
  Week 28 | -93.56 (8.382) | -81.47 (32.251) | -79.34 (28.091) | -66.53 (43.437) | -87.78 (13.648) | -74.18 (42.104) | -89.88 (6.304) | -74.54 (31.665) | -76.87 (31.377)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -86.08 (24.896) | -76.51 (38.401) | -69.06 (38.468) | -58.78 (44.767) | -91.07 (13.744) | -75.64 (41.038) | -93.76 (4.960) | -68.09 (34.850) | -71.98 (33.063)
  Week 36: number analyzed (Participants) | 13 | 33 | 10 | 28 | 12 | 32 | 7 | 32 | 15
  Week 36 | -86.56 (28.656) | -69.33 (43.838) | -66.64 (39.631) | -56.24 (46.469) | -91.22 (13.203) | -75.77 (40.984) | -93.09 (6.000) | -67.27 (40.162) | -74.93 (32.664)
  Week 40: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 32 | 7 | 31 | 15
  Week 40 | -84.74 (28.948) | -65.65 (44.932) | -68.31 (38.024) | -57.39 (47.379) | -90.68 (13.737) | -64.68 (64.041) | -95.55 (5.011) | -70.11 (37.802) | -74.05 (32.343)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -84.46 (28.757) | -66.73 (44.328) | -69.41 (38.731) | -56.30 (46.700) | -90.18 (12.912) | -62.46 (63.983) | -83.57 (21.909) | -69.98 (37.145) | -72.99 (33.353)
  Week 48: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -71.66 (40.416) | -65.18 (44.327) | -66.61 (39.645) | -53.59 (48.780) | -90.26 (12.961) | -57.47 (65.142) | -88.02 (22.234) | -66.63 (40.889) | -70.92 (33.888)
  Week 52: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 29 | 7 | 31 | 14
  Week 52 | -71.22 (40.152) | -61.78 (44.406) | -68.09 (37.719) | -53.58 (48.725) | -89.09 (15.625) | -54.42 (65.177) | -86.51 (22.331) | -69.76 (38.241) | -72.04 (34.827)

11. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in EASI (EASI 50) (Part 1)
Description: as for outcome 1
Time Frame: Baseline to weeks 2, 4, 8, 12, 16, 20 and 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. Participant with missing data were considered as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 2 | 19.5 | 15.4 | 16.9 | 22.8 | 13.9
  Week 4 | 29.9 | 21.8 | 39.0 | 39.2 | 24.1
  Week 8 | 45.5 | 38.5 | 53.2 | 54.4 | 27.8
  Week 12 | 62.3 | 44.9 | 61.0 | 62.0 | 26.6
  Week 16 | 63.6 | 52.6 | 57.1 | 65.8 | 27.8
  Week 20 | 63.6 | 51.3 | 58.4 | 58.2 | 25.3
  Week 24 | 66.2 | 43.6 | 55.8 | 53.2 | 24.1

12. Secondary Outcome: Percentage of Participants With at Least a 75% Reduction From Baseline in EASI (EASI 75) (Part 1)
Description: as for outcome 1
Time Frame: Baseline at weeks 2, 4, 8, 12, 16, 20 and 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to week 24. Participants with missing data were considered as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 2 | 9.1 | 2.6 | 2.6 | 2.5 | 5.1
  Week 4 | 9.1 | 9.0 | 11.7 | 11.4 | 6.3
  Week 8 | 23.4 | 16.7 | 27.3 | 25.3 | 8.9
  Week 12 | 33.8 | 25.6 | 44.2 | 43.0 | 11.4
  Week 16 | 40.3 | 38.5 | 42.9 | 40.5 | 11.4
  Week 20 | 49.4 | 42.3 | 48.1 | 40.5 | 13.9
  Week 24 | 54.5 | 38.5 | 49.4 | 40.5 | 17.7

13. Secondary Outcome: Percentage of Participants With at Least a 90% Reduction From Baseline in EASI (EASI 90) (Part 1)
Description: as for outcome 1
Time Frame: Baseline to weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 2 | 2.6 | 1.3 | 0 | 1.3 | 0
  Week 4 | 6.5 | 1.3 | 1.3 | 2.5 | 0
  Week 8 | 7.8 | 7.7 | 9.1 | 8.9 | 1.3
  Week 12 | 10.4 | 9.0 | 14.3 | 12.7 | 5.1
  Week 16 | 15.6 | 14.1 | 16.9 | 19.0 | 3.8
  Week 20 | 27.3 | 23.1 | 24.7 | 19.0 | 7.6
  Week 24 | 37.7 | 26.9 | 32.5 | 24.1 | 11.4

14. Secondary Outcome: Percentage of Participants With a 100% Reduction From Baseline in EASI (EASI 100) (Part 1)
Description: as for outcome 1
Time Frame: Baseline to weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 2 | 0 | 1.3 | 0 | 0 | 0
  Week 4 | 2.6 | 0 | 0 | 0 | 0
  Week 8 | 2.6 | 5.1 | 1.3 | 0 | 0
  Week 12 | 3.9 | 2.6 | 2.6 | 2.5 | 0
  Week 16 | 3.9 | 1.3 | 2.6 | 1.3 | 1.3
  Week 20 | 6.5 | 6.4 | 3.9 | 2.5 | 1.3
  Week 24 | 7.8 | 6.4 | 9.1 | 1.3 | 3.8

15. Secondary Outcome: Change in IGA (Investigator Global Assessment) From Baseline to (Week 24) (Part 1)
Description: The IGA is a five-point scale that provides a global clinical assessment of AD severity ranging from 0 to 4, where 0 indicates clear, 1 is almost clear, 2 is mild, 3 is moderate, and 4 indicates severe AD
Time Frame: Baseline to weeks 2, 4, 8, 12, 16, 20, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Score on a scale
  Week 2: number analyzed (Participants) | 73 | 77 | 75 | 75 | 78
  Week 2 | -0.33 (0.625) | -0.21 (0.408) | -0.29 (0.540) | -0.23 (0.481) | -0.18 (0.503)
  Week 4: number analyzed (Participants) | 76 | 74 | 76 | 77 | 75
  Week 4 | -0.57 (0.869) | -0.38 (0.590) | -0.45 (0.620) | -0.51 (0.661) | -0.31 (0.592)
  Week 8: number analyzed (Participants) | 70 | 70 | 75 | 76 | 72
  Week 8 | -0.79 (0.976) | -0.74 (0.829) | -0.80 (0.900) | -0.76 (0.709) | -0.32 (0.728)
  Week 12: number analyzed (Participants) | 70 | 70 | 72 | 77 | 70
  Week 12 | -1.10 (1.024) | -0.87 (0.867) | -1.04 (1.013) | -1.00 (0.973) | -0.36 (0.660)
  Week 16: number analyzed (Participants) | 70 | 69 | 73 | 76 | 69
  Week 16 | -1.23 (0.981) | -0.99 (0.899) | -0.96 (1.033) | -1.09 (0.969) | -0.43 (0.757)
  Week 20: number analyzed (Participants) | 67 | 69 | 72 | 72 | 67
  Week 20 | -1.43 (1.118) | -1.17 (1.137) | -1.11 (1.120) | -1.10 (0.981) | -0.45 (0.822)
  Week 24: number analyzed (Participants) | 71 | 68 | 72 | 70 | 67
  Week 24 | -1.48 (1.205) | -1.16 (1.241) | -1.32 (1.265) | -1.16 (1.030) | -0.49 (0.959)

16. Secondary Outcome: Change in IGA (Investigator Global Assessment) From Baseline (Part 2)
Description: as for outcome 15
Time Frame: Baseline to weeks 24, 28, 31, 36, 40, 44, 48 & 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (500 mg LD) at Part 1) were re-randomized to receive KY1005 250mg Q4W from Week 24 to Week 52
- Placebo Re-randomized From the 250mg (LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (500 mg LD) at Part 1) were re-randomized to receive placebo Q4W from Week 24 to Week 52
- 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (no LD) at Part 1) were rerandomized to receive KY1005 250mg Q4W from Week 24 to Week 52
- Placebo Re-randomized From the 250mg (No LD) Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 250 mg (no LD) at Part 1) were rerandomized to receive placebo Q4W from Week 24 to Week 52
- Placebo Re-randomized From the 125 mg Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 125 mg at Part 1) were rerandomized to receive placebo Q4W from Week 24 to Week 52
- 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (62.5 mg) were re-randomized to receive KY1005 62.5mg Q4W from Week 24 to Week 52
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Score on a scale
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 5 | 33 | 16
  Week 24 | -2.31 (0.855) | -1.91 (1.026) | -2.00 (0.953) | -1.82 (1.156) | -2.42 (0.793) | -1.82 (1.131) | -2.00 (1.000) | -1.73 (0.911) | -1.63 (1.204)
  Week 28: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 7 | 34 | 14
  Week 28 | -2.46 (0.967) | -2.00 (1.155) | -2.17 (1.193) | -1.46 (1.138) | -2.25 (0.965) | -1.74 (1.064) | -1.71 (0.951) | -1.47 (0.961) | -1.71 (1.383)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -2.00 (1.000) | -1.82 (1.314) | -1.73 (1.348) | -1.32 (1.188) | -2.33 (0.985) | -1.75 (1.078) | -1.71 (0.951) | -1.41 (1.160) | -1.67 (1.234)
  Week 36: number analyzed (Participants) | 13 | 33 | 10 | 28 | 12 | 32 | 7 | 32 | 15
  Week 36 | -2.08 (1.188) | -1.70 (1.380) | -1.40 (1.174) | -1.29 (1.182) | -2.17 (1.115) | -1.81 (1.230) | -2.00 (1.000) | -1.53 (1.344) | -1.67 (1.234)
  Week 40: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 32 | 7 | 31 | 15
  Week 40 | -2.08 (1.115) | -1.71 (1.395) | -1.64 (1.286) | -1.29 (1.301) | -2.36 (1.120) | -1.75 (1.164) | -1.86 (1.215) | -1.58 (1.311) | -1.53 (1.302)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -2.00 (1.155) | -1.69 (1.447) | -1.73 (1.348) | -1.32 (1.335) | -2.08 (1.084) | -1.63 (1.070) | -1.71 (1.113) | -1.58 (1.259) | -1.64 (1.393)
  Week 48: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -1.69 (1.182) | -1.69 (1.469) | -1.60 (1.350) | -1.36 (1.367) | -2.08 (1.240) | -1.50 (1.137) | -2.00 (1.414) | -1.63 (1.351) | -1.71 (1.590)
  Week 52: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 29 | 7 | 31 | 14
  Week 52 | -1.77 (1.301) | -1.55 (1.434) | -1.64 (1.286) | -1.36 (1.420) | -2.18 (1.401) | -1.48 (1.214) | -2.00 (1.155) | -1.65 (1.305) | -1.79 (1.672)

17. Secondary Outcome: Percentage of Participants With a Score of IGA (Investigator Global Assessment) 0 or 1 and a Reduction From Baseline of ≥ 2 Points (Part 1)
Description: The IGA is a five-point scale that provides a global clinical assessment of AD (Atopic Dermatitis) severity ranging from 0 to 4, where 0 indicates clear, 1 is almost clear, 2 is mild, 3 is moderate, and 4 indicates severe AD
Time Frame: Baseline to weeks 2, 4, 8,12,16,20 & 24
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 2 | 1.3 | 0 | 0 | 0 | 1.3
  Week 4 | 5.2 | 1.3 | 1.3 | 2.5 | 2.5
  Week 8 | 9.1 | 9.0 | 13.0 | 5.1 | 5.1
  Week 12 | 16.9 | 12.8 | 19.5 | 19.0 | 3.8
  Week 16 | 22.1 | 14.1 | 19.5 | 25.3 | 5.1
  Week 20 | 33.8 | 25.6 | 27.3 | 21.5 | 8.9
  Week 24 | 45.5 | 33.3 | 40.3 | 29.1 | 11.4

18. Secondary Outcome: Absolute Change in SCORAD (SCORing Atopic Dermatitis) Index From Baseline (Part 1)
Description: SCORAD was used to assess the extent and severity of AD (Atopic Dermatitis). Extent and severity of eczema as well as subjective assessment of symptoms were assessed and scored. SCORAD total score ranges from 0 (absent disease) to 103 (severe disease)
Time Frame: Baseline to weeks 4, 8, 12, 16, 20 & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Score on a scale
  Week 4: number analyzed (Participants) | 76 | 74 | 76 | 77 | 75
  Week 4 | -15.30 (16.517) | -12.27 (13.455) | -15.89 (14.865) | -14.43 (13.691) | -11.13 (14.243)
  Week 8: number analyzed (Participants) | 70 | 70 | 75 | 76 | 72
  Week 8 | -22.39 (19.368) | -19.61 (17.527) | -21.49 (19.200) | -21.42 (16.956) | -12.50 (16.584)
  Week 12: number analyzed (Participants) | 70 | 70 | 72 | 77 | 70
  Week 12 | -27.80 (19.621) | -22.31 (17.936) | -27.72 (20.084) | -26.45 (19.649) | -13.97 (16.898)
  Week 16: number analyzed (Participants) | 70 | 69 | 73 | 76 | 68
  Week 16 | -30.12 (20.086) | -25.07 (20.233) | -26.28 (21.258) | -28.15 (19.831) | -13.85 (18.123)
  Week 20: number analyzed (Participants) | 67 | 69 | 72 | 72 | 67
  Week 20 | -34.89 (22.369) | -28.04 (22.472) | -29.80 (23.594) | -26.71 (21.056) | -13.91 (19.325)
  Week 24: number analyzed (Participants) | 71 | 68 | 70 | 70 | 67
  Week 24 | -36.19 (24.605) | -27.28 (22.937) | -29.96 (25.735) | -28.48 (21.793) | -15.08 (22.739)

19. Secondary Outcome: Absolute Change in SCORAD (SCORing Atopic Dermatitis) Index From Baseline (Part 2)
Description: as for outcome 18
Time Frame: Baseline to week 24, 28, 32, 36, 40, 44, 48 & 52
Population: The Full Analysis Set (FAS2) for Part 2 included all re-randomized participants at week 24.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Placebo Re-randomized From the 125mg Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 125 mg at Part 1) were rerandomized to receive placebo Q4W from Week 24 to Week 52
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Score on a scale
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -52.22 (14.314) | -44.25 (21.373) | -42.44 (21.879) | -36.77 (21.919) | -49.87 (13.012) | -41.65 (24.173) | -45.20 (18.017) | -38.45 (22.077) | -40.54 (23.584)
  Week 28: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 7 | 34 | 13
  Week 28 | -54.19 (18.525) | -44.30 (23.737) | -43.38 (24.261) | -33.40 (23.845) | -47.15 (16.401) | -43.95 (24.475) | -41.17 (19.190) | -37.46 (23.843) | -42.98 (24.770)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -51.19 (23.086) | -41.55 (25.962) | -37.58 (27.000) | -28.31 (23.318) | -50.76 (16.285) | -44.04 (22.541) | -40.76 (17.685) | -36.72 (25.421) | -37.81 (25.964)
  Week 36: number analyzed (Participants) | 13 | 33 | 10 | 28 | 12 | 32 | 7 | 32 | 15
  Week 36 | -49.68 (25.709) | -38.72 (27.164) | -33.91 (26.686) | -27.91 (24.154) | -52.12 (19.167) | -45.28 (23.438) | -40.09 (16.767) | -37.15 (27.483) | -39.35 (25.340)
  Week 40: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 32 | 7 | 31 | 15
  Week 40 | -49.88 (26.342) | -38.96 (29.090) | -36.05 (27.550) | -30.05 (26.602) | -52.42 (19.560) | -42.93 (24.694) | -45.31 (22.710) | -37.75 (27.127) | -36.74 (25.865)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -47.38 (26.194) | -38.61 (28.602) | -37.95 (28.362) | -29.98 (26.387) | -51.14 (20.299) | -40.96 (24.470) | -36.39 (21.651) | -36.83 (27.061) | -37.47 (27.887)
  Week 48: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -39.75 (25.447) | -38.18 (29.948) | -35.13 (27.409) | -29.71 (28.021) | -52.40 (22.250) | -38.38 (24.940) | -43.80 (27.380) | -37.64 (28.543) | -38.10 (28.181)
  Week 52: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 29 | 7 | 30 | 14
  Week 52 | -40.26 (26.751) | -34.69 (28.925) | -35.04 (27.120) | -29.26 (27.488) | -50.26 (26.772) | -37.07 (25.763) | -42.26 (25.861) | -38.41 (26.915) | -39.94 (29.182)

20. Secondary Outcome: Percentage Change in SCORAD (SCORing Atopic Dermatitis) Index From Baseline (Part 1)
Description: as for outcome 18
Time Frame: Baseline to weeks 4, 8, 12, 16, 20, & 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of change
  Week 4: number analyzed (Participants) | 76 | 74 | 76 | 77 | 75
  Week 4 | -22.02 (22.050) | -18.52 (20.315) | -22.76 (20.903) | -21.42 (21.101) | -16.67 (21.045)
  Week 8: number analyzed (Participants) | 70 | 70 | 75 | 76 | 72
  Week 8 | -31.84 (24.549) | -30.00 (28.050) | -30.47 (26.260) | -32.07 (23.600) | -18.27 (23.875)
  Week 12: number analyzed (Participants) | 70 | 70 | 72 | 77 | 70
  Week 12 | -40.32 (25.145) | -33.64 (26.502) | -39.38 (27.228) | -39.22 (26.807) | -20.70 (24.587)
  Week 16: number analyzed (Participants) | 70 | 69 | 73 | 76 | 68
  Week 16 | -43.25 (26.555) | -37.18 (28.395) | -37.33 (29.071) | -41.44 (26.134) | -20.87 (26.791)
  Week 20: number analyzed (Participants) | 67 | 69 | 72 | 72 | 67
  Week 20 | -49.92 (28.279) | -42.07 (32.179) | -42.30 (32.422) | -39.05 (28.347) | -20.88 (28.527)
  Week 24: number analyzed (Participants) | 71 | 68 | 70 | 70 | 67
  Week 24 | -57.87 (32.609) | -41.04 (34.212) | -42.58 (35.812) | -41.49 (29.263) | -22.21 (33.233)

21. Secondary Outcome: Percentage Change in SCORAD (SCORing Atopic Dermatitis) Index From Baseline (Part 2)
Description: as for outcome 18
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48 & 52
Population: The Full Analysis Set (FAS2) for Part 2 included all re-randomized at week 24. Only those participants with data available at specified time points are reported.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of change
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -76.47 (11.581) | -63.86 (27.005) | -60.09 (26.373) | -57.73 (34.302) | -72.55 (15.422) | -58.96 (31.260) | -66.12 (19.532) | -55.75 (26.945) | -60.13 (33.848)
  Week 28: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 7 | 34 | 13
  Week 28 | -78.39 (16.236) | -63.35 (28.625) | -62.58 (32.229) | -52.12 (35.950) | -68.39 (21.143) | -61.69 (32.214) | -64.22 (18.649) | -53.98 (29.707) | -62.81 (36.300)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -72.44 (25.786) | -59.37 (33.889) | -53.42 (34.955) | -44.49 (35.890) | -74.03 (21.589) | -62.38 (31.104) | -64.07 (16.853) | -52.47 (31.788) | -56.11 (38.003)
  Week 36: number analyzed (Participants) | 13 | 33 | 10 | 28 | 12 | 32 | 7 | 32 | 15
  Week 36 | -71.50 (31.364) | -55.13 (35.598) | -49.88 (36.111) | -43.78 (36.278) | -75.08 (21.563) | -63.79 (31.710) | -64.24 (20.730) | -53.95 (35.053) | -58.72 (36.827)
  Week 40: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 32 | 7 | 31 | 15
  Week 40 | -71.43 (31.643) | -54.79 (38.533) | -51.85 (37.053) | -46.81 (39.055) | -74.34 (22.474) | -61.12 (34.217) | -70.27 (22.037) | -54.56 (34.785) | -54.24 (36.614)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -67.26 (31.749) | -54.96 (38.272) | -54.10 (37.251) | -46.95 (39.736) | -73.34 (22.409) | -57.94 (33.953) | -58.19 (33.365) | -52.89 (34.032) | -55.26 (39.204)
  Week 48: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -59.99 (35.979) | -53.71 (39.548) | -51.66 (37.347) | -45.48 (41.426) | -74.37 (23.066) | -54.55 (34.719) | -67.92 (35.766) | -54.29 (35.851) | -56.30 (39.696)
  Week 52: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 29 | 7 | 30 | 14
  Week 52 | -60.41 (36.686) | -49.90 (40.104) | -49.68 (35.129) | -44.93 (40.527) | -69.62 (29.104) | -52.47 (35.396) | -65.97 (34.709) | -56.19 (34.460) | -58.86 (40.701)

22. Secondary Outcome: Absolute Change in Affected Body Surface Area (BSA) From Baseline (Part 1)
Time Frame: Baseline to weeks 2, 4, 8, 12, 16, 20, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of body surface area
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of body surface area
  Week 2: number analyzed (Participants) | 32 | 36 | 36 | 39 | 38
  Week 2 | -4.50 (10.610) | -5.61 (10.165) | -9.08 (15.999) | -7.41 (12.588) | -4.84 (9.113)
  Week 4: number analyzed (Participants) | 76 | 74 | 76 | 77 | 75
  Week 4 | -12.83 (15.922) | -10.16 (12.917) | -13.34 (17.347) | -12.51 (16.318) | -9.67 (16.941)
  Week 8: number analyzed (Participants) | 70 | 70 | 75 | 76 | 72
  Week 8 | -19.37 (18.857) | -15.77 (17.004) | -17.55 (21.064) | -19.11 (18.253) | -10.00 (17.375)
  Week 12: number analyzed (Participants) | 70 | 70 | 72 | 77 | 70
  Week 12 | -24.13 (18.097) | -19.54 (19.578) | -21.94 (22.715) | -24.14 (19.903) | -11.46 (17.035)
  Week 16: number analyzed (Participants) | 70 | 69 | 73 | 76 | 68
  Week 16 | -26.91 (20.286) | -22.71 (21.966) | -21.74 (24.799) | -26.04 (20.403) | -8.87 (16.956)
  Week 20: number analyzed (Participants) | 67 | 69 | 72 | 72 | 67
  Week 20 | -30.25 (21.850) | -23.33 (22.600) | -24.35 (26.238) | -24.63 (21.263) | -11.04 (19.653)
  Week 24: number analyzed (Participants) | 71 | 68 | 70 | 70 | 67
  Week 24 | -31.35 (22.434) | -21.82 (21.882) | -22.66 (27.317) | -25.77 (22.085) | -10.45 (20.837)

23. Secondary Outcome: Absolute Change in Affected BSA From Baseline (Part 2)
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48 & 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percentage of body surface area
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of body surface area
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -46.92 (22.009) | -37.94 (18.723) | -37.17 (17.994) | -28.14 (21.790) | -41.17 (22.982) | -33.81 (26.454) | -40.60 (26.006) | -34.30 (19.787) | -32.06 (22.831)
  Week 28: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 7 | 34 | 13
  Week 28 | -48.69 (23.329) | -38.68 (20.582) | -35.92 (20.804) | -25.54 (22.718) | -40.00 (23.394) | -35.61 (25.720) | -37.14 (23.801) | -33.62 (19.692) | -36.00 (24.553)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -47.15 (25.271) | -36.62 (23.049) | -29.64 (25.590) | -23.21 (23.710) | -42.08 (22.685) | -35.94 (26.193) | -38.00 (23.847) | -32.13 (21.515) | -30.07 (22.861)
  Week 36: number analyzed (Participants) | 13 | 33 | 10 | 28 | 12 | 32 | 7 | 32 | 15
  Week 36 | -46.00 (26.242) | -33.61 (24.187) | -28.30 (26.437) | -22.21 (23.857) | -41.67 (23.051) | -35.75 (25.664) | -37.86 (24.674) | -30.91 (24.288) | -31.27 (24.391)
  Week 40: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 32 | 7 | 31 | 15
  Week 40 | -46.62 (26.314) | -32.94 (24.589) | -29.18 (24.774) | -22.57 (23.841) | -41.45 (23.729) | -33.41 (22.649) | -39.57 (24.758) | -32.00 (23.697) | -31.27 (24.566)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -47.23 (26.540) | -33.22 (24.143) | -29.73 (25.503) | -22.21 (23.706) | -42.17 (25.283) | -31.91 (22.069) | -34.43 (25.172) | -32.23 (23.250) | -27.43 (20.478)
  Week 48: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -35.69 (26.183) | -32.72 (25.358) | -28.30 (26.378) | -21.50 (24.053) | -42.92 (25.336) | -30.53 (23.544) | -36.43 (21.141) | -31.13 (26.208) | -26.93 (20.775)
  Week 52: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 29 | 7 | 30 | 14
  Week 52 | -35.54 (26.384) | -29.48 (22.232) | -29.55 (25.359) | -21.46 (23.562) | -45.09 (25.770) | -29.66 (23.818) | -34.71 (18.688) | -33.33 (22.702) | -27.21 (20.955)

24. Secondary Outcome: Percentage Change in Affected BSA From Baseline (Part 1)
Time Frame: Baseline to weeks 2, 4, 8, 12, 16, 20, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage change
  Week 2: number analyzed (Participants) | 32 | 36 | 36 | 39 | 38
  Week 2 | -10.11 (24.013) | -12.23 (26.053) | -19.43 (30.139) | -15.06 (37.312) | -11.45 (22.767)
  Week 4: number analyzed (Participants) | 76 | 74 | 76 | 77 | 75
  Week 4 | -26.45 (28.733) | -23.44 (28.941) | -29.46 (32.934) | -28.84 (38.412) | -20.92 (38.260)
  Week 8: number analyzed (Participants) | 70 | 70 | 75 | 76 | 72
  Week 8 | -39.12 (31.915) | -36.01 (35.268) | -37.60 (36.988) | -42.84 (33.931) | -21.24 (40.914)
  Week 12: number analyzed (Participants) | 70 | 70 | 72 | 77 | 70
  Week 12 | -49.88 (29.737) | -43.68 (38.140) | -47.04 (40.519) | -52.16 (35.736) | -26.56 (36.705)
  Week 16: number analyzed (Participants) | 70 | 69 | 73 | 76 | 68
  Week 16 | -54.58 (32.206) | -49.44 (40.861) | -46.35 (43.511) | -56.36 (35.593) | -22.37 (40.483)
  Week 20: number analyzed (Participants) | 67 | 69 | 72 | 72 | 67
  Week 20 | -59.75 (33.804) | -51.07 (42.023) | -50.36 (45.871) | -53.55 (42.762) | -25.46 (42.034)
  Week 24: number analyzed (Participants) | 71 | 68 | 70 | 70 | 67
  Week 24 | -63.02 (36.184) | -49.42 (43.012) | -48.11 (48.748) | -52.94 (44.872) | -23.76 (44.394)

25. Secondary Outcome: Percentage Change in Affected BSA From Baseline (Part 2)
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48 & 52
Population: The Full Analysis Set (FAS2) for Part 2 included all re-randomized participants at week 24. Only those participants with data available at specified time points are reported.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage change
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -88.09 (12.983) | -78.75 (27.966) | -80.67 (27.843) | -67.85 (39.902) | -85.29 (19.008) | -71.05 (39.900) | -80.52 (14.717) | -74.02 (31.419) | -72.91 (34.317)
  Week 28: number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 31 | 7 | 34 | 13
  Week 28 | -90.51 (10.816) | -79.51 (29.501) | -76.55 (35.680) | -62.09 (42.748) | -81.75 (24.996) | -73.28 (40.454) | -88.57 (5.800) | -72.98 (30.947) | -75.14 (37.955)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -83.58 (23.940) | -75.09 (36.907) | -65.07 (49.743) | -55.89 (45.768) | -86.34 (18.724) | -74.61 (40.429) | -90.31 (10.263) | -66.90 (35.357) | -69.74 (38.644)
  Week 36: number analyzed (Participants) | 13 | 33 | 10 | 28 | 12 | 32 | 7 | 32 | 15
  Week 36 | -81.56 (27.924) | -68.81 (40.261) | -61.93 (51.222) | -53.48 (45.933) | -85.33 (18.348) | -74.73 (40.570) | -89.70 (10.552) | -63.85 (46.152) | -72.34 (39.621)
  Week 40: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 32 | 7 | 31 | 15
  Week 40 | -82.62 (28.019) | -66.33 (41.876) | -64.54 (49.422) | -54.92 (47.035) | -86.81 (17.237) | -72.10 (41.016) | -94.09 (5.083) | -66.00 (43.207) | -72.08 (39.691)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -83.52 (28.118) | -66.91 (41.122) | -65.39 (49.945) | -53.82 (46.414) | -84.47 (24.104) | -69.38 (41.133) | -81.11 (19.107) | -66.54 (41.241) | -70.30 (40.560)
  Week 48: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -69.37 (40.195) | -64.74 (42.092) | -62.01 (51.359) | -52.52 (47.479) | -85.70 (19.040) | -64.73 (42.700) | -87.79 (16.209) | -62.58 (48.827) | -68.01 (40.428)
  Week 52: number analyzed (Participants) | 13 | 31 | 11 | 28 | 11 | 29 | 7 | 30 | 14
  Week 52 | -68.90 (40.301) | -61.59 (42.339) | -64.90 (49.605) | -52.82 (47.733) | -89.06 (14.176) | -62.25 (42.451) | -85.46 (16.921) | -68.75 (39.935) | -68.78 (41.236)

26. Secondary Outcome: Absolute Change in Patient Oriented Eczema Measure (POEM) From Baseline (Part 1)
Description: POEM is a 7-item (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) questionnaire to assess frequency of disease symptoms with a scoring system of 0 to 28. The higher score indicating higher severity
Time Frame: Baseline to weeks 4, 8, 12, 16, 20, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Score on a scale
  Week 4: number analyzed (Participants) | 75 | 74 | 76 | 77 | 75
  Week 4 | -4.40 (6.403) | -4.01 (6.287) | -5.42 (6.498) | -4.08 (5.448) | -2.32 (5.910)
  Week 8: number analyzed (Participants) | 70 | 70 | 74 | 76 | 72
  Week 8 | -7.03 (6.869) | -5.13 (7.093) | -5.70 (6.943) | -6.75 (6.646) | -2.13 (6.400)
  Week 12: number analyzed (Participants) | 69 | 70 | 72 | 77 | 70
  Week 12 | -7.87 (7.286) | -6.50 (7.229) | -7.29 (7.216) | -7.36 (7.460) | -2.26 (6.088)
  Week 16: number analyzed (Participants) | 69 | 69 | 73 | 76 | 68
  Week 16 | -8.28 (7.286) | -7.23 (7.744) | -7.19 (7.720) | -7.32 (7.017) | -2.37 (6.867)
  Week 20: number analyzed (Participants) | 66 | 69 | 72 | 72 | 67
  Week 20 | -9.39 (7.577) | -7.13 (8.662) | -8.10 (8.150) | -7.39 (7.721) | -2.33 (6.821)
  Week 24: number analyzed (Participants) | 70 | 68 | 70 | 70 | 67
  Week 24 | -9.96 (7.888) | -7.21 (8.213) | -7.86 (8.572) | -7.64 (7.011) | -2.19 (7.310)

27. Secondary Outcome: Absolute Change in Patient Oriented Eczema Measure (POEM) From Baseline (Part 2)
Description: as for outcome 26
Time Frame: Baseline to weeks 24, 32, 36, 40, 44, 48 & 52
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Score on a scale
  Week 24: number analyzed (Participants) | 13 | 33 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -15.31 (6.061) | -11.97 (6.410) | -11.58 (8.586) | -9.25 (8.347) | -11.75 (7.086) | -10.42 (7.580) | -14.00 (6.205) | -9.45 (7.155) | -8.75 (7.197)
  Week 32: number analyzed (Participants) | 13 | 30 | 11 | 28 | 12 | 31 | 7 | 31 | 13
  Week 32 | -14.69 (8.499) | -10.23 (8.320) | -11.91 (8.240) | -6.79 (8.875) | -12.83 (7.082) | -11.32 (8.113) | -11.29 (10.323) | -9.42 (7.784) | -7.62 (8.856)
  Week 36: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 32 | 7 | 32 | 14
  Week 36 | -13.23 (8.738) | -9.91 (8.129) | -11.90 (7.264) | -7.00 (8.932) | -13.00 (7.019) | -11.75 (8.370) | -12.57 (9.502) | -8.66 (7.790) | -7.93 (7.966)
  Week 40: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 32 | 7 | 31 | 14
  Week 40 | -13.92 (8.411) | -9.10 (8.715) | -11.00 (6.633) | -7.82 (9.302) | -11.73 (8.162) | -11.88 (8.698) | -11.29 (8.995) | -8.81 (8.300) | -7.50 (7.714)
  Week 44: number analyzed (Participants) | 13 | 31 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -13.31 (8.460) | -9.81 (8.920) | -10.45 (6.699) | -6.50 (8.804) | -11.92 (8.262) | -10.19 (8.361) | -7.86 (7.515) | -8.71 (8.158) | -7.93 (7.908)
  Week 48: number analyzed (Participants) | 13 | 31 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -11.69 (9.861) | -10.39 (8.519) | -11.50 (6.916) | -7.50 (9.268) | -11.75 (9.836) | -10.33 (8.125) | -9.57 (9.126) | -9.90 (8.660) | -7.50 (8.438)
  Week 52: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 29 | 7 | 31 | 14
  Week 52 | -11.85 (10.148) | -9.13 (8.320) | -11.36 (6.889) | -6.82 (9.318) | -10.64 (10.053) | -8.55 (8.240) | -10.00 (9.452) | -8.58 (9.164) | -8.50 (9.146)

28. Secondary Outcome: Percentage Change in Patient Oriented Eczema Measure (POEM) From Baseline (Part 1)
Description: as for outcome 26
Time Frame: Baseline to weeks 4, 8, 12, 16, 20, & 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of change
  Week 4: number analyzed (Participants) | 75 | 73 | 76 | 77 | 75
  Week 4 | -20.81 (34.179) | -21.02 (31.360) | -22.77 (30.783) | -17.94 (30.152) | -8.99 (39.554)
  Week 8: number analyzed (Participants) | 70 | 69 | 74 | 76 | 72
  Week 8 | -33.06 (41.272) | -26.52 (33.397) | -26.62 (34.946) | -34.60 (31.584) | -6.28 (42.851)
  Week 12: number analyzed (Participants) | 69 | 69 | 72 | 77 | 70
  Week 12 | -36.22 (43.169) | -32.42 (32.145) | -33.33 (33.732) | -34.61 (34.275) | -8.04 (41.445)
  Week 16: number analyzed (Participants) | 69 | 68 | 73 | 76 | 68
  Week 16 | -37.08 (52.391) | -34.71 (34.574) | -32.78 (36.449) | -35.49 (32.862) | -8.12 (45.515)
  Week 20: number analyzed (Participants) | 66 | 68 | 72 | 72 | 67
  Week 20 | -44.03 (38.850) | -34.23 (38.938) | -37.38 (38.448) | -35.37 (36.589) | -8.32 (44.942)
  Week 24: number analyzed (Participants) | 70 | 67 | 70 | 70 | 67
  Week 24 | -44.69 (61.808) | -33.91 (48.273) | -36.65 (40.947) | -36.81 (34.444) | -6.98 (49.837)

29. Secondary Outcome: Percentage Change in Patient Oriented Eczema Measure (POEM) From Baseline (Part 2)
Description: as for outcome 26
Time Frame: Baseline to weeks 24, 32, 36, 40. 44, 48, & 52
Population: The Full Analysis Set (FAS2) for Part 2 included all re-randomized participants at week 24. Only those participants with data available at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of change
  Week 24: number analyzed (Participants) | 13 | 33 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -72.61 (19.898) | -61.00 (30.657) | -54.05 (38.147) | -46.08 (37.356) | -60.03 (30.545) | -51.61 (35.438) | -64.00 (20.049) | -45.63 (34.579) | -47.92 (40.572)
  Week 32: number analyzed (Participants) | 13 | 30 | 11 | 28 | 12 | 31 | 7 | 31 | 13
  Week 32 | -64.90 (38.029) | -50.03 (44.543) | -56.00 (35.875) | -30.61 (39.689) | -64.21 (28.981) | -55.82 (36.229) | -47.30 (57.463) | -46.42 (38.011) | -43.95 (50.962)
  Week 36: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 32 | 7 | 32 | 14
  Week 36 | -60.09 (40.508) | -48.61 (43.883) | -57.09 (34.068) | -33.73 (38.724) | -66.78 (27.084) | -57.38 (37.436) | -57.54 (59.987) | -43.35 (40.000) | -44.58 (45.387)
  Week 40: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 32 | 7 | 31 | 14
  Week 40 | -62.85 (38.659) | -44.35 (45.524) | -54.47 (35.815) | -37.89 (40.032) | -58.98 (33.289) | -58.12 (38.754) | -49.79 (55.862) | -43.75 (40.933) | -42.88 (45.567)
  Week 44: number analyzed (Participants) | 13 | 31 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -60.83 (40.648) | -48.48 (47.524) | -52.24 (36.218) | -30.25 (43.110) | -59.17 (35.572) | -50.10 (37.814) | -36.09 (53.637) | -43.16 (39.688) | -46.19 (46.429)
  Week 48: number analyzed (Participants) | 13 | 31 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -54.56 (46.380) | -51.53 (44.857) | -55.93 (35.043) | -35.37 (42.309) | -58.18 (46.077) | -51.56 (39.299) | -44.04 (58.904) | -50.45 (41.809) | -43.48 (48.292)
  Week 52: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 29 | 7 | 31 | 14
  Week 52 | -54.68 (45.987) | -44.51 (43.725) | -54.47 (34.319) | -29.38 (46.373) | -52.64 (47.556) | -43.45 (42.459) | -48.82 (63.478) | -43.01 (45.577) | -47.62 (50.785)

30. Secondary Outcome: Absolute Change in Dermatology Life Quality Index (DLQI) From Baseline (Parts 1)
Description: DLQI is a questionnaire with a score system of 0 to 30 the high score is indicative of poor QoL.
Time Frame: Baseline to weeks 2, 8, 16, 20, & 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Score on a scale
  Week 2: number analyzed (Participants) | 71 | 77 | 75 | 75 | 78
  Week 2 | -3.63 (4.992) | -2.82 (4.850) | -3.32 (5.745) | -3.40 (5.131) | -2.09 (4.710)
  Week 8: number analyzed (Participants) | 70 | 69 | 74 | 76 | 72
  Week 8 | -6.13 (6.164) | -5.59 (5.553) | -5.08 (7.252) | -7.13 (5.954) | -2.43 (5.466)
  Week 16: number analyzed (Participants) | 67 | 67 | 73 | 76 | 68
  Week 16 | -7.79 (6.832) | -6.25 (6.246) | -6.47 (7.835) | -7.76 (6.265) | -2.35 (6.069)
  Week 20: number analyzed (Participants) | 66 | 69 | 72 | 72 | 67
  Week 20 | -7.89 (6.848) | -6.42 (6.833) | -6.97 (8.512) | -7.31 (7.132) | -2.39 (6.391)
  Week 24: number analyzed (Participants) | 70 | 68 | 70 | 70 | 67
  Week 24 | -8.33 (7.036) | -6.54 (6.384) | -6.74 (8.681) | -7.69 (7.230) | -2.30 (6.406)

31. Secondary Outcome: Absolute Change in Dermatology Life Quality Index (DLQI) From Baseline (Part 2)
Description: DLQI is a questionnaire with a score system of 0 to 30 the high score is indicative of poor QoL.
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48, & 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Placebo Re-randomized From the 62.5mg Arm (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) (who received 62.5 mg at Part 1) were rerandomized to receive placebo Q4W from Week 24 to Week 52
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Score on a scale
  Week 24: number analyzed (Participants) | 13 | 33 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -12.54 (6.703) | -9.00 (6.290) | -9.08 (6.487) | -7.57 (7.295) | -11.42 (7.115) | -8.26 (9.338) | -15.40 (8.562) | -9.67 (7.712) | -6.44 (7.420)
  Week 28: number analyzed (Participants) | 13 | 33 | 12 | 28 | 12 | 31 | 7 | 34 | 13
  Week 28 | -12.62 (8.191) | -9.52 (6.929) | -9.83 (6.658) | -7.21 (6.488) | -11.33 (7.832) | -8.45 (9.705) | -12.29 (9.232) | -9.68 (8.029) | -5.77 (8.633)
  Week 32: number analyzed (Participants) | 13 | 33 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -12.38 (8.272) | -8.00 (7.612) | -8.55 (8.238) | -5.75 (7.183) | -12.25 (7.700) | -8.50 (9.629) | -13.14 (8.050) | -9.13 (7.906) | -5.47 (7.963)
  Week 36: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 32 | 7 | 32 | 14
  Week 36 | -11.85 (8.122) | -7.72 (7.985) | -7.90 (6.903) | -6.18 (7.222) | -12.58 (7.716) | -8.84 (9.893) | -14.00 (8.446) | -8.53 (7.927) | -5.93 (7.839)
  Week 40: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 32 | 7 | 31 | 14
  Week 40 | -12.23 (7.715) | -7.07 (8.073) | -7.18 (5.456) | -6.21 (7.279) | -11.27 (7.976) | -8.06 (9.844) | -14.57 (7.569) | -8.23 (8.281) | -5.36 (8.308)
  Week 44: number analyzed (Participants) | 13 | 31 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -11.38 (8.109) | -7.19 (7.943) | -8.18 (6.258) | -5.68 (7.029) | -12.08 (8.426) | -6.88 (9.587) | -10.29 (7.889) | -8.26 (8.058) | -5.93 (6.889)
  Week 48: number analyzed (Participants) | 13 | 31 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -9.92 (6.800) | -7.29 (8.022) | -8.40 (7.516) | -6.21 (7.218) | -11.92 (8.229) | -6.83 (9.322) | -11.29 (6.237) | -7.93 (7.891) | -6.79 (7.040)
  Week 52: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 29 | 7 | 31 | 14
  Week 52 | -9.08 (6.652) | -6.83 (7.852) | -8.09 (7.077) | -5.93 (7.383) | -12.55 (9.136) | -6.41 (9.428) | -11.57 (6.705) | -8.10 (7.752) | -6.64 (6.902)

32. Secondary Outcome: Percentage Change in Dermatology Life Quality Index (DLQI) From Baseline (Part 1)
Description: DLQI is a questionnaire with a score system of 0 to 30 the high score is indicative of poor QoL.
Time Frame: Baseline to weeks 2, 8, 16, 20, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of change
  Week 2: number analyzed (Participants) | 71 | 77 | 75 | 74 | 78
  Week 2 | -22.68 (31.305) | -11.95 (47.921) | -16.80 (41.680) | -22.73 (32.711) | -10.30 (37.999)
  Week 8: number analyzed (Participants) | 70 | 69 | 74 | 75 | 72
  Week 8 | -36.87 (36.954) | -36.14 (41.176) | -27.54 (59.199) | -45.85 (32.198) | -13.12 (42.775)
  Week 16: number analyzed (Participants) | 67 | 67 | 73 | 75 | 68
  Week 16 | -46.69 (40.563) | -41.27 (43.616) | -34.02 (62.565) | -48.96 (29.801) | -11.35 (51.739)
  Week 20: number analyzed (Participants) | 66 | 69 | 72 | 72 | 67
  Week 20 | -47.48 (40.616) | -42.90 (46.336) | -35.79 (67.398) | -44.33 (36.816) | -12.08 (49.973)
  Week 24: number analyzed (Participants) | 70 | 68 | 70 | 70 | 67
  Week 24 | -51.84 (41.442) | -42.36 (45.550) | -33.28 (72.816) | -45.63 (33.860) | -11.91 (55.694)

33. Secondary Outcome: Percentage Change in Dermatology Life Quality Index (DLQI) From Baseline (Part 2)
Description: DLQI is a questionnaire with a score system of 0 to 30 the high score is indicative of poor QoL.
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48, & 52
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of change
  Week 24: number analyzed (Participants) | 13 | 33 | 12 | 28 | 12 | 31 | 5 | 33 | 16
  Week 24 | -75.53 (26.705) | -61.64 (35.809) | -64.74 (31.091) | -44.26 (57.217) | -72.47 (27.818) | -47.08 (82.439) | -70.77 (27.653) | -55.36 (33.443) | -48.30 (57.726)
  Week 28: number analyzed (Participants) | 13 | 33 | 12 | 28 | 12 | 31 | 7 | 34 | 13
  Week 28 | -72.50 (37.184) | -62.65 (43.216) | -71.77 (29.970) | -44.81 (56.575) | -70.02 (28.760) | -48.86 (83.936) | -65.28 (26.807) | -55.62 (34.382) | -41.13 (80.192)
  Week 32: number analyzed (Participants) | 13 | 33 | 11 | 28 | 12 | 32 | 7 | 32 | 15
  Week 32 | -68.19 (38.039) | -48.69 (56.833) | -61.68 (42.315) | -31.65 (55.087) | -77.14 (26.277) | -50.15 (83.141) | -72.98 (17.074) | -52.99 (36.735) | -41.18 (68.097)
  Week 36: number analyzed (Participants) | 13 | 32 | 10 | 28 | 12 | 32 | 7 | 32 | 14
  Week 36 | -65.76 (35.792) | -48.12 (56.610) | -60.50 (41.018) | -35.86 (58.071) | -79.13 (24.980) | -52.16 (84.141) | -78.26 (23.932) | -49.48 (43.137) | -45.04 (65.630)
  Week 40: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 32 | 7 | 31 | 14
  Week 40 | -69.26 (34.172) | -44.78 (59.798) | -58.29 (42.112) | -36.52 (58.909) | -72.31 (27.268) | -46.41 (84.277) | -83.18 (16.284) | -49.75 (42.024) | -38.69 (80.196)
  Week 44: number analyzed (Participants) | 13 | 31 | 11 | 28 | 12 | 32 | 7 | 31 | 14
  Week 44 | -63.03 (41.237) | -45.33 (60.470) | -63.04 (42.005) | -33.25 (58.480) | -76.32 (31.166) | -39.27 (83.804) | -60.44 (28.925) | -49.15 (43.228) | -48.21 (48.871)
  Week 48: number analyzed (Participants) | 13 | 31 | 10 | 28 | 12 | 30 | 7 | 30 | 14
  Week 48 | -59.02 (36.676) | -45.68 (59.933) | -63.97 (43.622) | -35.98 (57.915) | -73.10 (28.704) | -40.20 (84.240) | -70.04 (26.437) | -50.82 (41.018) | -57.92 (45.339)
  Week 52: number analyzed (Participants) | 13 | 30 | 11 | 28 | 11 | 29 | 7 | 31 | 14
  Week 52 | -53.62 (36.496) | -43.64 (56.804) | -61.04 (42.716) | -33.21 (59.514) | -72.35 (33.768) | -35.27 (85.953) | -71.56 (28.287) | -49.24 (43.003) | -57.12 (44.899)

34. Secondary Outcome: Absolute Change in Atopic Dermatitis Control Tool (ADCT) From Baseline (Part 1)
Description: ADCT is a questionnaire to assess patient-self-perceived control of their eczema with a total score from 0 to 24; higher scores indicate lower AD control
Time Frame: Baseline to weeks 16, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Score on a scale
  Week 16: number analyzed (Participants) | 67 | 66 | 73 | 76 | 68
  Week 16 | -6.70 (5.813) | -5.41 (6.054) | -6.22 (6.272) | -6.61 (5.804) | -2.50 (4.589)
  Week 24: number analyzed (Participants) | 65 | 66 | 70 | 68 | 67
  Week 24 | -7.35 (6.695) | -5.80 (6.187) | -6.70 (6.566) | -6.66 (5.868) | -1.90 (5.046)

35. Secondary Outcome: Absolute Change in Atopic Dermatitis Control Tool (ADCT) From Baseline (Part 2)
Description: as for outcome 34
Time Frame: Baseline to weeks 24, 36 & 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Score on a scale
  Week 24: number analyzed (Participants) | 13 | 28 | 12 | 27 | 12 | 31 | 5 | 31 | 16
  Week 24 | -11.23 (6.071) | -8.64 (5.927) | -9.83 (6.506) | -7.44 (5.673) | -9.83 (5.132) | -8.42 (6.386) | -12.60 (6.986) | -8.29 (5.996) | -6.25 (6.083)
  Week 36: number analyzed (Participants) | 13 | 30 | 10 | 27 | 12 | 31 | 7 | 31 | 13
  Week 36 | -11.46 (5.681) | -8.13 (6.463) | -8.20 (6.143) | -7.78 (6.123) | -10.33 (5.483) | -9.26 (6.875) | -10.71 (6.550) | -8.03 (6.385) | -6.38 (6.063)
  Week 52: number analyzed (Participants) | 13 | 30 | 11 | 27 | 11 | 29 | 7 | 29 | 14
  Week 52 | -11.31 (4.768) | -8.30 (5.706) | -8.82 (6.809) | -7.44 (6.594) | -10.45 (5.989) | -6.48 (6.539) | -9.71 (4.751) | -8.34 (6.893) | -7.14 (6.125)

36. Secondary Outcome: Percentage Change in Atopic Dermatitis Control Tool (ADCT) From Baseline (Part 1)
Description: as for outcome 34
Time Frame: Baseline to weeks 16, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of change
  Week 16: number analyzed (Participants) | 67 | 66 | 73 | 76 | 68
  Week 16 | -40.56 (37.340) | -33.42 (34.745) | -36.42 (37.103) | -38.72 (30.762) | -17.04 (32.553)
  Week 24: number analyzed (Participants) | 65 | 66 | 70 | 68 | 67
  Week 24 | -45.18 (42.438) | -36.20 (41.363) | -40.45 (40.708) | -39.35 (31.799) | -12.31 (37.504)

37. Secondary Outcome: Percentage Change in Atopic Dermatitis Control Tool (ADCT) From Baseline (Part 2)
Description: as for outcome 34
Time Frame: Baseline to weeks 24, 36 & 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of change
  Week 24: number analyzed (Participants) | 13 | 28 | 12 | 27 | 12 | 31 | 5 | 31 | 16
  Week 24 | -66.75 (32.632) | -57.08 (37.656) | -56.01 (36.112) | -49.97 (34.078) | -65.46 (26.823) | -53.10 (40.207) | -63.92 (29.784) | -50.66 (33.458) | -44.95 (45.331)
  Week 36: number analyzed (Participants) | 13 | 30 | 10 | 27 | 12 | 31 | 7 | 31 | 13
  Week 36 | -69.01 (29.493) | -50.38 (42.649) | -50.01 (37.199) | -50.87 (33.197) | -69.73 (28.925) | -58.44 (43.340) | -62.63 (23.130) | -48.59 (38.274) | -49.42 (45.902)
  Week 52: number analyzed (Participants) | 13 | 30 | 11 | 27 | 11 | 29 | 7 | 29 | 14
  Week 52 | -69.93 (26.250) | -54.77 (34.128) | -52.75 (41.167) | -47.15 (39.681) | -67.84 (32.469) | -41.39 (43.875) | -64.19 (28.274) | -50.29 (41.341) | -53.35 (47.196)

38. Secondary Outcome: Absolute Change in Hospital Anxiety and Depression Scale (HADS) From Baseline (Part 1)
Description: The HADS is 14-item questionnaire with two subscales: anxiety & depression. Each subscale (anxiety & depression) ranges 0-21. The total HADS score ranges 0-42 with higher score indicating a poorer state.
Time Frame: Baseline to weeks 8 16, 20, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Score on a scale
  Week 8: number analyzed (Participants) | 70 | 68 | 74 | 76 | 72
  Week 8 | -2.20 (4.639) | -2.07 (6.194) | -2.35 (5.641) | -3.29 (5.132) | -0.97 (3.940)
  Week 16: number analyzed (Participants) | 67 | 66 | 73 | 76 | 68
  Week 16 | -2.67 (5.761) | -2.53 (6.510) | -3.04 (6.292) | -3.74 (6.401) | -0.57 (5.088)
  Week 20: number analyzed (Participants) | 66 | 68 | 72 | 72 | 67
  Week 20 | -2.52 (7.254) | -2.35 (7.326) | -3.38 (6.787) | -4.24 (5.873) | -0.66 (4.176)
  Week 24: number analyzed (Participants) | 70 | 67 | 70 | 70 | 67
  Week 24 | -2.96 (7.550) | -2.30 (6.880) | -2.83 (6.818) | -4.00 (6.802) | -0.97 (4.196)

39. Secondary Outcome: Absolute Change in Hospital Anxiety and Depression Scale (HADS) From Baseline (Part 2)
Description: as for outcome 38
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48 & 52
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
score on a scale
  Week 24: number analyzed (Participants) | 13 | 33 | 12 | 27 | 12 | 31 | 5 | 33 | 16
  Week 24 | -4.54 (8.482) | -1.73 (7.434) | -5.58 (10.184) | -2.81 (6.822) | -3.67 (6.998) | -4.42 (7.890) | -8.20 (6.340) | -4.03 (6.710) | -0.38 (4.660)
  Week 28: number analyzed (Participants) | 13 | 33 | 12 | 27 | 12 | 31 | 7 | 34 | 13
  Week 28 | -3.54 (7.965) | -2.52 (6.205) | -6.50 (11.430) | -2.70 (6.916) | -4.33 (7.679) | -4.97 (8.428) | -7.29 (5.251) | -5.26 (7.034) | 0.38 (4.753)
  Week 32: number analyzed (Participants) | 13 | 33 | 11 | 27 | 12 | 32 | 7 | 32 | 15
  Week 32 | -3.38 (8.893) | -1.24 (6.996) | -4.09 (9.027) | -2.74 (7.593) | -4.42 (7.242) | -5.66 (8.280) | -6.86 (5.460) | -3.97 (6.483) | -0.20 (4.491)
  Week 36: number analyzed (Participants) | 13 | 32 | 10 | 27 | 12 | 32 | 7 | 32 | 14
  Week 36 | -1.85 (9.754) | -1.22 (8.015) | -3.80 (10.497) | -2.52 (5.833) | -4.42 (6.999) | -5.50 (8.828) | -7.14 (4.880) | -3.75 (7.878) | 0.29 (4.250)
  Week 40: number analyzed (Participants) | 13 | 30 | 11 | 27 | 11 | 32 | 7 | 31 | 14
  Week 40 | -2.92 (8.864) | -1.40 (6.966) | -3.09 (10.222) | -2.70 (6.151) | -3.55 (7.594) | -5.16 (8.674) | -7.43 (5.563) | -3.29 (5.593) | 0.50 (5.125)
  Week 44: number analyzed (Participants) | 13 | 31 | 11 | 27 | 12 | 32 | 7 | 31 | 14
  Week 44 | -2.69 (8.873) | -0.29 (6.963) | -3.45 (10.511) | -3.07 (5.313) | -4.25 (7.225) | -4.56 (8.879) | -5.43 (5.192) | -3.71 (7.408) | -0.21 (4.318)
  Week 48: number analyzed (Participants) | 13 | 31 | 10 | 27 | 12 | 30 | 7 | 30 | 14
  Week 48 | -3.08 (8.883) | -0.68 (7.078) | -4.40 (10.024) | -2.85 (5.559) | -3.33 (7.797) | -5.23 (8.724) | -7.43 (5.412) | -4.17 (7.269) | -1.00 (4.852)
  Week 52: number analyzed (Participants) | 13 | 30 | 11 | 27 | 11 | 29 | 7 | 31 | 14
  Week 52 | -2.46 (9.162) | -0.80 (7.092) | -2.55 (8.359) | -3.00 (5.877) | -4.18 (7.167) | -4.59 (8.454) | -7.29 (5.794) | -3.13 (8.082) | -0.64 (5.719)

40. Secondary Outcome: Percentage Change in Hospital Anxiety and Depression Scale (HADS) From Baseline (Part 1)
Description: as for outcome 38
Time Frame: Baseline to weeks 8, 16, 20, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of change
  Week 8: number analyzed (Participants) | 69 | 66 | 70 | 76 | 69
  Week 8 | -18.40 (46.151) | -11.76 (48.829) | -10.22 (56.395) | -13.15 (69.427) | -0.66 (77.969)
  Week 16: number analyzed (Participants) | 66 | 65 | 69 | 76 | 65
  Week 16 | -18.12 (56.175) | -11.72 (54.678) | -15.84 (54.001) | -17.47 (94.346) | 2.82 (101.930)
  Week 20: number analyzed (Participants) | 65 | 66 | 68 | 72 | 64
  Week 20 | -20.15 (65.506) | -7.39 (62.693) | -17.62 (59.518) | -25.97 (83.249) | -5.02 (78.180)
  Week 24: number analyzed (Participants) | 69 | 65 | 66 | 70 | 64
  Week 24 | -13.22 (97.953) | -8.67 (60.563) | -17.75 (52.049) | -12.07 (120.061) | -8.17 (77.872)

41. Secondary Outcome: Percentage Change in Hospital Anxiety and Depression Scale (HADS) From Baseline (Part 2)
Description: as for outcome 38
Time Frame: Baseline to weeks 24, 28, 32, 36, 40, 44, 48 & 52
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of change
  Week 24: number analyzed (Participants) | 13 | 32 | 11 | 26 | 11 | 29 | 5 | 33 | 16
  Week 24 | -28.01 (54.369) | -17.89 (76.693) | -34.27 (48.841) | -13.63 (65.697) | -20.28 (49.825) | -32.24 (65.070) | -46.94 (22.063) | -22.38 (58.898) | -32.55 (66.184)
  Week 28: number analyzed (Participants) | 13 | 32 | 11 | 26 | 11 | 29 | 7 | 34 | 13
  Week 28 | -18.57 (53.870) | -22.56 (67.645) | -30.97 (51.945) | -17.92 (53.098) | 4.22 (96.782) | -30.52 (66.305) | -49.58 (31.509) | -33.17 (41.412) | -38.39 (77.030)
  Week 32: number analyzed (Participants) | 13 | 32 | 10 | 26 | 11 | 30 | 7 | 32 | 15
  Week 32 | -19.06 (60.844) | -14.02 (82.893) | -29.10 (52.035) | -20.31 (63.189) | -11.36 (87.084) | -43.96 (68.306) | -42.56 (27.759) | -32.62 (49.764) | -38.06 (69.176)
  Week 36: number analyzed (Participants) | 13 | 31 | 9 | 26 | 11 | 30 | 7 | 32 | 14
  Week 36 | 11.76 (84.979) | -9.44 (81.662) | -6.28 (62.772) | -22.30 (51.020) | -8.75 (85.214) | -37.19 (71.372) | -51.27 (29.960) | -32.59 (49.531) | -9.11 (110.289)
  Week 40: number analyzed (Participants) | 13 | 29 | 10 | 26 | 10 | 30 | 7 | 31 | 14
  Week 40 | -13.29 (60.249) | -18.23 (79.025) | 7.25 (82.513) | -21.32 (50.659) | 4.24 (91.941) | -40.11 (67.991) | -56.66 (33.879) | -35.92 (46.888) | -1.02 (98.096)
  Week 44: number analyzed (Participants) | 13 | 30 | 10 | 26 | 11 | 30 | 7 | 31 | 14
  Week 44 | -2.42 (54.527) | -5.30 (88.418) | -23.23 (56.824) | -31.88 (49.100) | -15.90 (85.382) | -30.93 (71.891) | -41.44 (37.143) | -32.73 (57.357) | -22.21 (80.062)
  Week 48: number analyzed (Participants) | 13 | 30 | 9 | 26 | 11 | 28 | 7 | 30 | 14
  Week 48 | -14.15 (60.660) | -4.47 (95.509) | -28.27 (51.499) | -21.89 (53.010) | 4.97 (88.017) | -39.36 (69.672) | -60.77 (35.190) | -36.32 (47.746) | -34.95 (67.833)
  Week 52: number analyzed (Participants) | 13 | 29 | 10 | 26 | 11 | 28 | 7 | 31 | 14
  Week 52 | -8.10 (67.182) | -7.59 (92.868) | -13.70 (44.085) | -19.98 (56.405) | 0.43 (85.522) | -14.22 (78.739) | -59.23 (37.434) | -23.84 (50.933) | -18.16 (69.310)

42. Secondary Outcome: Absolute Change in Weekly Average of Pruritus Numerical Rating Scale (NRS) From Baseline (Part 1)
Description: as for outcome 5
Time Frame: Baseline to weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
score on a scale
  Week 1: number analyzed (Participants) | 74 | 77 | 77 | 77 | 77
  Week 1 | -0.54 (1.096) | -0.56 (0.978) | -0.49 (0.965) | -0.45 (0.908) | -0.28 (1.071)
  Week 2: number analyzed (Participants) | 75 | 77 | 76 | 76 | 77
  Week 2 | -0.65 (1.316) | -0.79 (1.367) | -0.73 (1.075) | -0.81 (1.224) | -0.42 (1.046)
  Week 3: number analyzed (Participants) | 75 | 77 | 77 | 77 | 76
  Week 3 | -0.90 (1.619) | -0.92 (1.392) | -1.05 (1.302) | -0.88 (1.478) | -0.65 (1.567)
  Week 4: number analyzed (Participants) | 75 | 76 | 76 | 77 | 77
  Week 4 | -.096 (1.672) | -1.25 (1.657) | -1.36 (1.443) | -1.09 (1.668) | -0.77 (1.744)
  Week 5: number analyzed (Participants) | 75 | 75 | 75 | 77 | 74
  Week 5 | -0.99 (1.811) | -1.38 (1.653) | -1.42 (1.591) | -1.49 (1.799) | -0.83 (2.030)
  Week 6: number analyzed (Participants) | 74 | 73 | 75 | 76 | 75
  Week 6 | -1.09 (1.679) | -1.35 (1.818) | -1.38 (1.666) | -1.58 (2.057) | -0.94 (1.899)
  Week 7: number analyzed (Participants) | 73 | 72 | 74 | 76 | 73
  Week 7 | -1.25 (1.966) | -1.54 (1.850) | -1.57 (1.710) | -1.78 (2.002) | -0.78 (1.922)
  Week 8: number analyzed (Participants) | 73 | 72 | 73 | 75 | 73
  Week 8 | -1.42 (2.062) | -1.50 (1.786) | -1.60 (1.816) | -1.93 (2.053) | -0.80 (1.979)
  Week 9: number analyzed (Participants) | 74 | 73 | 74 | 75 | 70
  Week 9 | -1.44 (2.104) | -1.52 (1.805) | -1.89 (1.885) | -2.13 (2.031) | -1.00 (2.142)
  Week 10: number analyzed (Participants) | 72 | 73 | 72 | 74 | 69
  Week 10 | -1.62 (2.162) | -1.67 (1.852) | -1.82 (2.082) | -2.17 (2.137) | -0.97 (2.244)
  Week 11: number analyzed (Participants) | 73 | 70 | 73 | 74 | 68
  Week 11 | -1.68 (2.176) | -1.67 (1.936) | -2.06 (2.091) | -2.31 (2.248) | -0.93 (2.111)
  Week 12: number analyzed (Participants) | 72 | 69 | 71 | 73 | 68
  Week 12 | -1.70 (2.204) | -1.65 (2.074) | -1.96 (2.107) | -2.28 (2.262) | -0.79 (2.162)
  Week 13: number analyzed (Participants) | 72 | 71 | 71 | 73 | 70
  Week 13 | -1.83 (2.295) | -1.87 (2.247) | -2.05 (2.164) | -2.28 (2.291) | -0.72 (2.087)
  Week 14: number analyzed (Participants) | 72 | 70 | 70 | 75 | 67
  Week 14 | -1.82 (2.355) | -2.02 (2.468) | -2.13 (2.308) | -2.35 (2.316) | -0.58 (2.055)
  Week 15: number analyzed (Participants) | 70 | 69 | 71 | 74 | 67
  Week 15 | -1.87 (2.386) | -2.08 (2.511) | -2.10 (2.290) | -2.32 (2.288) | -0.57 (2.018)
  Week 16: number analyzed (Participants) | 72 | 68 | 71 | 75 | 66
  Week 16 | -2.06 (2.539) | -2.09 (2.497) | -2.22 (2.275) | -2.31 (2.301) | -0.54 (2.077)
  Week 17: number analyzed (Participants) | 70 | 68 | 71 | 75 | 67
  Week 17 | -2.13 (2.465) | -2.18 (2.457) | -2.14 (2.368) | -2.35 (2.346) | -0.61 (2.143)
  Week 18: number analyzed (Participants) | 70 | 68 | 68 | 75 | 66
  Week 18 | -2.18 (2.534) | -2.21 (2.543) | -2.16 (2.307) | -2.37 (2.383) | -0.55 (2.168)
  Week 19: number analyzed (Participants) | 69 | 67 | 70 | 75 | 67
  Week 19 | -2.19 (2.484) | -2.22 (2.563) | -2.14 (2.291) | -2.38 (2.463) | -0.75 (2.278)
  Week 20: number analyzed (Participants) | 68 | 67 | 69 | 72 | 67
  Week 20 | -2.28 (2.522) | -2.19 (2.530) | -2.13 (2.360) | -2.31 (2.401) | -0.67 (2.201)
  Week 21: number analyzed (Participants) | 69 | 68 | 70 | 72 | 67
  Week 21 | -2.28 (2.516) | -2.23 (2.576) | -2.27 (2.352) | -2.43 (2.404) | -0.76 (2.332)
  Week 22: number analyzed (Participants) | 69 | 66 | 69 | 72 | 67
  Week 22 | -2.38 (2.622) | -2.29 (2.699) | -2.25 (2.438) | -2.44 (2.383) | -0.73 (2.314)
  Week 23: number analyzed (Participants) | 70 | 67 | 70 | 71 | 67
  Week 23 | -2.56 (2.671) | -2.27 (2.538) | -2.20 (2.529) | -2.59 (2.453) | -0.61 (2.215)
  Week 24: number analyzed (Participants) | 70 | 66 | 70 | 71 | 67
  Week 24 | -2.58 (2.662) | -2.30 (2.672) | -2.21 (2.616) | -2.46 (2.427) | -0.55 (2.224)

43. Secondary Outcome: Absolute Change in Weekly Average of Pruritus Numerical Rating Scale (NRS) From Baseline (Part 2)
Description: as for outcome 5
Time Frame: Baseline to weeks 24, 25, 26, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 38, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, 51, & 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 250 mg KY1005 Re-randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Score on a scale
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 26 | 11 | 33 | 6 | 33 | 16
  Week 24 | -3.63 (2.380) | -2.83 (2.909) | -4.00 (2.711) | -2.25 (2.861) | -4.34 (2.169) | -2.92 (2.539) | -4.63 (1.822) | -2.82 (2.571) | -1.95 (3.083)
  Week 25: number analyzed (Participants) | 13 | 34 | 12 | 25 | 12 | 31 | 6 | 33 | 15
  Week 25 | -3.83 (2.353) | -2.73 (2.973) | -4.08 (2.726) | -2.42 (2.895) | -4.12 (2.413) | -2.81 (2.405) | -4.92 (1.863) | -2.64 (2.577) | -2.08 (3.177)
  Week 26: number analyzed (Participants) | 13 | 33 | 12 | 25 | 11 | 30 | 7 | 33 | 15
  Week 26 | -3.82 (2.442) | -2.71 (2.891) | -3.75 (2.654) | -2.33 (3.096) | -3.83 (2.428) | -2.56 (2.400) | -4.56 (1.903) | -2.70 (2.634) | -1.93 (3.202)
  Week 27: number analyzed (Participants) | 13 | 33 | 12 | 24 | 11 | 30 | 7 | 33 | 14
  Week 27 | -3.84 (2.444) | -2.58 (2.819) | -3.65 (2.619) | -2.28 (2.994) | -4.09 (2.567) | -2.84 (2.467) | -4.51 (1.790) | -2.57 (2.748) | -2.04 (3.351)
  Week 28: number analyzed (Participants) | 13 | 33 | 12 | 26 | 11 | 31 | 7 | 32 | 14
  Week 28 | -3.86 (2.432) | -2.56 (2.892) | -3.59 (2.575) | -2.29 (2.782) | -4.02 (2.525) | -3.01 (2.504) | -4.38 (1.827) | -2.75 (2.753) | -1.89 (3.459)
  Week 29: number analyzed (Participants) | 13 | 32 | 11 | 25 | 12 | 31 | 7 | 31 | 14
  Week 29 | -3.73 (2.612) | -2.51 (2.874) | -3.81 (2.425) | -1.85 (2.733) | -4.16 (2.387) | -2.99 (2.591) | -4.50 (2.035) | -2.64 (2.695) | -1.81 (3.386)
  Week 30: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 31 | 6 | 32 | 13
  Week 30 | -3.32 (2.564) | -2.78 (3.030) | -3.76 (2.394) | -2.07 (2.564) | -4.44 (2.526) | -2.68 (2.490) | -3.73 (2.125) | -2.59 (2.653) | -1.80 (3.445)
  Week 31: number analyzed (Participants) | 13 | 32 | 11 | 26 | 12 | 31 | 6 | 33 | 15
  Week 31 | -3.41 (2.580) | -2.74 (3.213) | -3.73 (2.431) | -1.71 (2.980) | -4.18 (2.428) | -2.81 (2.662) | -4.02 (2.280) | -2.78 (2.691) | -1.46 (3.132)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 25 | 12 | 32 | 7 | 33 | 14
  Week 32 | -3.43 (2.607) | -2.56 (3.098) | -3.13 (2.818) | -1.51 (2.736) | -4.27 (2.261) | -2.86 (2.617) | -4.40 (2.170) | -2.68 (2.674) | -1.54 (3.221)
  Week 33: number analyzed (Participants) | 13 | 34 | 11 | 26 | 12 | 32 | 7 | 33 | 14
  Week 33 | -3.60 (2.722) | -2.49 (3.220) | -3.06 (2.755) | -1.85 (2.867) | -4.32 (2.316) | -2.83 (2.579) | -4.14 (1.843) | -2.66 (2.705) | -1.45 (3.332)
  Week 34: number analyzed (Participants) | 13 | 33 | 11 | 26 | 12 | 31 | 7 | 32 | 13
  Week 34 | -3.49 (2.644) | -2.26 (3.114) | -3.32 (2.732) | -1.30 (2.792) | -4.43 (2.297) | -2.84 (2.508) | -3.97 (1.948) | -2.58 (2.665) | -1.86 (3.578)
  Week 35: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 32 | 7 | 31 | 14
  Week 35 | -3.47 (2.712) | -2.51 (3.219) | -3.09 (2.600) | -1.42 (2.685) | -4.60 (2.497) | -3.01 (2.529) | -4.55 (2.055) | -2.65 (2.674) | -1.86 (3.390)
  Week 36: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 32 | 7 | 30 | 14
  Week 36 | -3.48 (2.752) | -2.47 (3.262) | -2.81 (2.693) | -1.64 (2.670) | -4.67 (2.468) | -2.90 (2.527) | -4.14 (1.845) | -2.39 (2.626) | -1.56 (3.318)
  Week 37: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 31 | 7 | 30 | 14
  Week 37 | -3.44 (2.726) | -2.53 (3.244) | -2.50 (2.523) | -1.85 (2.758) | -4.51 (2.429) | -3.11 (2.508) | -4.49 (1.992) | -2.33 (2.564) | -1.58 (3.328)
  Week 38: number analyzed (Participants) | 13 | 33 | 11 | 26 | 12 | 32 | 7 | 30 | 13
  Week 38 | -3.31 (3.182) | -2.33 (3.159) | -2.06 (2.464) | -1.74 (2.803) | -4.57 (2.505) | -3.16 (2.672) | -4.52 (2.046) | -2.37 (2.548) | -1.64 (3.449)
  Week 39: number analyzed (Participants) | 13 | 32 | 11 | 26 | 12 | 32 | 7 | 29 | 14
  Week 39 | -3.34 (3.206) | -2.35 (3.212) | -2.52 (2.462) | -1.81 (2.792) | -4.24 (2.451) | -3.07 (2.548) | -4.66 (2.070) | -2.27 (2.605) | -1.78 (3.350)
  Week 40: number analyzed (Participants) | 13 | 32 | 10 | 26 | 12 | 32 | 6 | 29 | 14
  Week 40 | -3.29 (3.245) | -2.26 (3.208) | -2.11 (2.064) | -1.74 (2.697) | -4.24 (2.419) | -2.92 (2.574) | -2.98 (1.946) | -2.38 (2.659) | -1.67 (3.413)
  Week 41: number analyzed (Participants) | 13 | 32 | 9 | 26 | 12 | 31 | 7 | 29 | 13
  Week 41 | -3.25 (3.188) | -2.26 (3.213) | -1.82 (1.991) | -1.97 (2.774) | -4.56 (2.344) | -2.67 (2.798) | -3.73 (2.142) | -2.41 (2.697) | -1.64 (3.856)
  Week 42: number analyzed (Participants) | 13 | 32 | 11 | 27 | 12 | 32 | 7 | 30 | 13
  Week 42 | -3.21 (3.218) | -2.28 (3.307) | -2.53 (2.603) | -1.91 (2.835) | -4.67 (2.494) | -2.92 (2.876) | -3.78 (2.183) | -2.24 (2.655) | -2.01 (3.719)
  Week 43: number analyzed (Participants) | 13 | 32 | 11 | 27 | 12 | 32 | 7 | 30 | 12
  Week 43 | -3.30 (3.246) | -2.27 (3.158) | -2.53 (2.523) | -1.74 (2.821) | -4.64 (2.864) | -2.82 (2.612) | -3.70 (2.063) | -2.22 (2.736) | -2.31 (3.823)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 27 | 12 | 32 | 7 | 30 | 13
  Week 44 | -3.34 (3.276) | -2.31 (3.196) | -2.37 (2.349) | -1.79 (2.690) | -4.83 (2.484) | -2.81 (2.693) | -3.51 (2.084) | -2.21 (2.656) | -2.01 (3.730)
  Week 45: number analyzed (Participants) | 12 | 32 | 10 | 27 | 12 | 31 | 7 | 30 | 13
  Week 45 | -3.63 (3.034) | -2.41 (3.267) | -1.97 (2.110) | -1.87 (2.745) | -4.68 (2.637) | -2.62 (2.636) | -3.58 (1.992) | -2.23 (2.678) | -1.87 (3.752)
  Week 46: number analyzed (Participants) | 12 | 32 | 10 | 27 | 12 | 31 | 7 | 29 | 11
  Week 46 | -3.29 (3.359) | -2.46 (3.219) | -2.61 (2.550) | -1.84 (2.679) | -4.41 (2.864) | -2.33 (2.614) | -3.78 (2.146) | -2.28 (2.713) | -1.99 (4.071)
  Week 47: number analyzed (Participants) | 12 | 32 | 9 | 27 | 12 | 31 | 7 | 30 | 13
  Week 47 | -3.17 (3.283) | -2.31 (3.183) | -1.95 (2.320) | -1.84 (2.796) | -4.46 (2.830) | -2.30 (2.731) | -3.66 (2.139) | -2.38 (2.645) | -1.78 (3.762)
  Week 48: number analyzed (Participants) | 12 | 32 | 9 | 27 | 12 | 30 | 7 | 29 | 13
  Week 48 | -2.82 (3.247) | -2.43 (3.202) | -2.36 (2.366) | -1.84 (2.761) | -4.64 (2.892) | -2.04 (2.636) | -3.96 (2.251) | -2.31 (2.731) | -2.05 (3.716)
  Week 49: number analyzed (Participants) | 12 | 31 | 10 | 27 | 12 | 30 | 7 | 30 | 12
  Week 49 | -2.80 (3.230) | -2.27 (3.139) | -2.66 (2.610) | -2.02 (2.909) | -4.68 (2.893) | -2.02 (2.625) | -3.65 (1.938) | -2.46 (2.847) | -2.06 (3.875)
  Week 50: number analyzed (Participants) | 12 | 31 | 10 | 27 | 12 | 29 | 7 | 30 | 12
  Week 50 | -2.78 (3.223) | -2.23 (3.218) | -2.44 (2.699) | -1.90 (2.913) | -4.56 (2.923) | -1.87 (2.596) | -3.78 (2.092) | -2.35 (2.788) | -2.16 (3.870)
  Week 51: number analyzed (Participants) | 12 | 30 | 10 | 27 | 11 | 29 | 7 | 30 | 12
  Week 51 | -2.67 (3.188) | -2.42 (3.317) | -2.39 (2.399) | -1.80 (2.860) | -4.64 (3.094) | -1.89 (2.692) | -3.66 (2.014) | -2.40 (2.777) | -2.12 (3.883)
  Week 52: number analyzed (Participants) | 12 | 30 | 9 | 27 | 12 | 29 | 7 | 30 | 12
  Week 52 | -2.70 (3.119) | -2.17 (3.152) | -2.53 (2.917) | -1.84 (2.779) | -4.74 (2.909) | -1.84 (2.929) | -3.86 (2.135) | -2.33 (2.811) | -2.12 (3.904)

44. Secondary Outcome: Percent Change in Weekly Average of Pruritus Numerical Rating Scale (NRS) From Baseline (Part 1)
Description: as for outcome 5
Time Frame: Baseline to weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 & 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of change
  Week 1: number analyzed (Participants) | 74 | 77 | 77 | 77 | 77
  Week 1 | -6.26 (16.312) | -7.25 (13.575) | -6.18 (13.809) | -6.05 (13.049) | -3.70 (16.432)
  Week 2: number analyzed (Participants) | 75 | 77 | 76 | 76 | 77
  Week 2 | -7.50 (20.644) | -10.37 (19.307) | -9.86 (14.734) | -11.20 (18.124) | -5.63 (15.340)
  Week 3: number analyzed (Participants) | 75 | 77 | 77 | 77 | 76
  Week 3 | -11.08 (24.712) | -12.11 (18.977) | -14.11 (17.784) | -12.08 (22.244) | -7.89 (22.004)
  Week 4: number analyzed (Participants) | 75 | 76 | 76 | 77 | 77
  Week 4 | -12.16 (25.287) | -16.73 (22.997) | -18.37 (19.932) | -14.95 (24.356) | -9.83 (24.266)
  Week 5: number analyzed (Participants) | 75 | 75 | 75 | 77 | 74
  Week 5 | -12.58 (27.613) | -18.64 (23.725) | -19.20 (21.900) | -20.17 (25.112) | -10.14 (29.071)
  Week 6: number analyzed (Participants) | 74 | 73 | 75 | 76 | 75
  Week 6 | -13.73 (25.374) | -17.59 (25.814) | -18.68 (22.790) | -21.29 (28.179) | -12.43 (27.184)
  Week 7: number analyzed (Participants) | 73 | 72 | 74 | 76 | 73
  Week 7 | -15.89 (28.992) | -20.18 (25.476) | -21.18 (23.816) | -24.03 (27.650) | -10.18 (28.308)
  Week 8: number analyzed (Participants) | 73 | 72 | 73 | 75 | 73
  Week 8 | -18.41 (31.375) | -19.99 (24.992) | -21.14 (24.981) | -26.10 (27.810) | -10.51 (29.803)
  Week 9: number analyzed (Participants) | 74 | 73 | 74 | 75 | 70
  Week 9 | -18.83 (32.003) | -20.36 (25.407) | -25.45 (24.895) | -29.18 (27.455) | -13.34 (32.225)
  Week 10: number analyzed (Participants) | 72 | 73 | 72 | 74 | 69
  Week 10 | -21.19 (32.110) | -22.53 (25.815) | -24.46 (28.280) | -29.43 (28.109) | -12.99 (33.194)
  Week 11: number analyzed (Participants) | 73 | 70 | 73 | 74 | 68
  Week 11 | -21.93 (31.966) | -22.37 (26.321) | -27.67 (28.079) | -31.26 (29.641) | -12.73 (31.638)
  Week 12: number analyzed (Participants) | 72 | 69 | 71 | 73 | 68
  Week 12 | -22.59 (32.927) | -22.05 (28.445) | -26.52 (28.426) | -31.23 (30.323) | -10.62 (32.707)
  Week 13: number analyzed (Participants) | 72 | 71 | 71 | 73 | 70
  Week 13 | -23.88 (33.561) | -24.71 (30.761) | -28.18 (29.401) | -31.36 (31.724) | -10.05 (32.122)
  Week 14: number analyzed (Participants) | 72 | 70 | 70 | 75 | 67
  Week 14 | -23.87 (34.926) | -26.45 (32.870) | -29.19 (30.904) | -32.57 (31.719) | -7.60 (31.351)
  Week 15: number analyzed (Participants) | 70 | 69 | 71 | 74 | 67
  Week 15 | -24.40 (34.899) | -27.46 (33.838) | -28.87 (31.207) | -32.01 (30.980) | -6.87 (29.583)
  Week 16: number analyzed (Participants) | 72 | 68 | 71 | 75 | 66
  Week 16 | -26.85 (36.332) | -27.92 (33.619) | -30.75 (30.460) | -31.97 (31.194) | -6.62 (30.591)
  Week 17: number analyzed (Participants) | 70 | 68 | 71 | 75 | 67
  Week 17 | -27.81 (35.262) | -29.27 (33.331) | -29.68 (31.753) | -32.60 (31.851) | -7.46 (31.529)
  Week 18: number analyzed (Participants) | 70 | 68 | 68 | 75 | 66
  Week 18 | -28.78 (36.738) | -29.49 (34.514) | -29.89 (31.200) | -32.50 (32.096) | -6.37 (31.752)
  Week 19: number analyzed (Participants) | 69 | 67 | 70 | 75 | 67
  Week 19 | -28.98 (36.372) | -29.78 (35.087) | -29.83 (31.632) | -32.77 (33.698) | -9.50 (33.411)
  Week 20: number analyzed (Participants) | 68 | 67 | 69 | 72 | 67
  Week 20 | -30.61 (37.215) | -29.30 (34.365) | -29.48 (32.361) | -31.85 (32.767) | -8.56 (32.725)
  Week 21: number analyzed (Participants) | 69 | 68 | 70 | 72 | 67
  Week 21 | -30.40 (36.928) | -29.63 (34.869) | -31.61 (32.551) | -33.20 (33.098) | -9.71 (34.201)
  Week 22: number analyzed (Participants) | 69 | 66 | 69 | 72 | 67
  Week 22 | -31.81 (38.100) | -30.35 (36.881) | -31.15 (33.763) | -33.28 (32.108) | -9.36 (34.161)
  Week 23: number analyzed (Participants) | 70 | 67 | 70 | 71 | 67
  Week 23 | -34.26 (38.693) | -30.30 (35.236) | -30.52 (35.354) | -35.25 (33.102) | -7.23 (32.486)
  Week 24: number analyzed (Participants) | 70 | 66 | 70 | 71 | 67
  Week 24 | -34.70 (38.656) | -30.44 (36.696) | -30.64 (36.647) | -33.26 (32.433) | -6.66 (32.550)

45. Secondary Outcome: Percent Change in Weekly Average of Pruritus Numerical Rating Scale (NRS) From Baseline (Part 2)
Description: as for outcome 5
Time Frame: as for outcome 43
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | 250 mg KY1005 Re-randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Percentage of change
  Week 24: number analyzed (Participants) | 13 | 34 | 12 | 26 | 11 | 33 | 6 | 33 | 16
  Week 24 | -49.61 (33.036) | -38.71 (44.259) | -52.36 (33.258) | -29.76 (40.611) | -56.60 (24.568) | -42.27 (36.685) | -59.49 (22.140) | -38.95 (34.963) | -29.09 (44.653)
  Week 25: number analyzed (Participants) | 13 | 34 | 12 | 25 | 12 | 31 | 6 | 33 | 15
  Week 25 | -52.15 (31.579) | -36.78 (45.402) | -53.26 (33.810) | -31.69 (40.647) | -54.31 (29.223) | -41.26 (34.643) | -63.84 (23.417) | -37.04 (36.046) | -30.81 (46.001)
  Week 26: number analyzed (Participants) | 13 | 33 | 12 | 25 | 11 | 30 | 7 | 33 | 15
  Week 26 | -51.62 (32.197) | -36.84 (44.342) | -48.88 (32.071) | -30.68 (42.883) | -50.31 (29.134) | -38.14 (35.393) | -57.52 (22.280) | -37.71 (37.451) | -28.48 (46.252)
  Week 27: number analyzed (Participants) | 13 | 33 | 12 | 24 | 11 | 30 | 7 | 33 | 14
  Week 27 | -52.09 (32.613) | -35.34 (44.056) | -47.36 (30.909) | -29.42 (40.379) | -53.62 (30.255) | -42.65 (36.665) | -57.00 (20.810) | -35.32 (38.963) | -29.92 (48.506)
  Week 28: number analyzed (Participants) | 13 | 33 | 12 | 26 | 11 | 31 | 7 | 32 | 14
  Week 28 | -52.36 (32.642) | -34.80 (45.063) | -47.19 (31.551) | -30.58 (38.398) | -53.08 (30.684) | -44.86 (36.493) | -56.28 (24.247) | -38.37 (38.703) | -27.74 (49.936)
  Week 29: number analyzed (Participants) | 13 | 32 | 11 | 25 | 12 | 31 | 7 | 31 | 14
  Week 29 | -50.48 (35.634) | -34.13 (44.735) | -50.29 (29.286) | -24.35 (38.746) | -54.93 (28.705) | -44.31 (37.579) | -56.79 (23.453) | -36.46 (38.211) | -26.40 (48.994)
  Week 30: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 31 | 6 | 32 | 13
  Week 30 | -44.79 (34.219) | -37.91 (46.288) | -49.35 (28.435) | -28.00 (35.916) | -58.70 (30.600) | -40.30 (37.098) | -48.05 (24.892) | -36.03 (38.742) | -26.58 (49.832)
  Week 31: number analyzed (Participants) | 13 | 32 | 11 | 26 | 12 | 31 | 6 | 33 | 15
  Week 31 | -46.03 (34.355) | -37.18 (49.311) | -49.01 (28.581) | -21.78 (41.439) | -55.77 (30.420) | -42.26 (39.161) | -52.67 (29.311) | -39.45 (38.697) | -21.51 (44.331)
  Week 32: number analyzed (Participants) | 13 | 34 | 11 | 25 | 12 | 32 | 7 | 33 | 14
  Week 32 | -46.40 (35.233) | -34.68 (47.719) | -40.69 (34.523) | -19.61 (37.935) | -57.32 (29.140) | -42.64 (38.113) | -56.51 (27.668) | -37.63 (38.453) | -22.64 (46.122)
  Week 33: number analyzed (Participants) | 13 | 34 | 11 | 26 | 12 | 32 | 7 | 33 | 14
  Week 33 | -48.66 (36.625) | -33.52 (48.881) | -39.31 (33.036) | -24.61 (39.502) | -57.76 (29.406) | -42.45 (38.100) | -52.89 (22.337) | -37.50 (39.368) | -21.49 (48.348)
  Week 34: number analyzed (Participants) | 13 | 33 | 11 | 26 | 12 | 31 | 7 | 32 | 13
  Week 34 | -47.09 (35.098) | -30.56 (48.227) | -43.33 (34.277) | -17.18 (39.855) | -59.41 (29.414) | -42.96 (37.718) | -50.34 (22.937) | -35.63 (37.586) | -27.22 (51.629)
  Week 35: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 32 | 7 | 31 | 14
  Week 35 | -46.67 (36.047) | -33.99 (48.416) | -40.21 (32.239) | -18.51 (37.670) | -61.70 (32.381) | -44.99 (37.080) | -58.12 (24.772) | -36.74 (37.592) | -27.11 (48.897)
  Week 36: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 32 | 7 | 30 | 14
  Week 36 | -46.63 (36.326) | -33.43 (48.720) | -36.23 (33.872) | -22.43 (37.322) | -62.54 (31.831) | -43.37 (37.251) | -52.78 (22.120) | -33.66 (38.520) | -22.57 (47.897)
  Week 37: number analyzed (Participants) | 13 | 34 | 11 | 27 | 12 | 31 | 7 | 30 | 14
  Week 37 | -45.95 (35.161) | -34.42 (48.542) | -32.60 (31.909) | -25.63 (39.489) | -60.49 (31.510) | -46.52 (37.336) | -58.05 (27.565) | -33.22 (38.367) | -22.63 (48.038)
  Week 38: number analyzed (Participants) | 13 | 33 | 11 | 26 | 12 | 32 | 7 | 30 | 13
  Week 38 | -43.12 (42.814) | -31.62 (47.534) | -26.80 (31.244) | -24.20 (40.063) | -60.83 (31.559) | -47.17 (39.147) | -58.43 (27.410) | -33.72 (37.516) | -24.07 (49.645)
  Week 39: number analyzed (Participants) | 13 | 32 | 11 | 26 | 12 | 32 | 7 | 29 | 14
  Week 39 | -43.54 (42.937) | -31.75 (48.313) | -32.75 (31.185) | -25.49 (40.126) | -56.79 (31.763) | -46.10 (38.082) | -59.36 (25.162) | -32.70 (38.945) | -25.98 (48.229)
  Week 40: number analyzed (Participants) | 13 | 32 | 10 | 26 | 12 | 32 | 6 | 29 | 14
  Week 40 | -42.94 (43.748) | -30.52 (48.657) | -27.37 (25.233) | -24.24 (38.972) | -56.78 (31.397) | -43.62 (38.048) | -38.57 (22.074) | -34.20 (39.168) | -24.22 (49.044)
  Week 41: number analyzed (Participants) | 13 | 32 | 9 | 26 | 12 | 31 | 7 | 29 | 13
  Week 41 | -42.33 (43.065) | -30.85 (48.900) | -22.99 (23.218) | -27.38 (39.966) | -61.18 (30.487) | -39.66 (42.054) | -47.95 (26.092) | -34.51 (40.123) | -24.13 (55.219)
  Week 42: number analyzed (Participants) | 13 | 32 | 11 | 27 | 12 | 32 | 7 | 30 | 13
  Week 42 | -41.68 (42.874) | -30.76 (50.332) | -34.23 (35.319) | -26.33 (40.513) | -62.53 (32.149) | -42.91 (42.866) | -49.33 (29.448) | -32.01 (39.405) | -29.48 (53.423)
  Week 43: number analyzed (Participants) | 13 | 32 | 11 | 27 | 12 | 32 | 7 | 30 | 12
  Week 43 | -42.86 (43.495) | -30.51 (48.200) | -33.86 (33.053) | -23.93 (40.455) | -62.27 (36.647) | -41.66 (38.115) | -48.09 (26.148) | -31.34 (41.919) | -33.70 (54.865)
  Week 44: number analyzed (Participants) | 13 | 32 | 11 | 27 | 12 | 32 | 7 | 30 | 13
  Week 44 | -43.47 (44.000) | -31.71 (49.607) | -31.76 (30.960) | -24.67 (37.725) | -64.61 (31.787) | -42.36 (40.085) | -46.04 (28.399) | -31.28 (40.103) | -29.07 (53.672)
  Week 45: number analyzed (Participants) | 12 | 32 | 10 | 27 | 12 | 31 | 7 | 30 | 13
  Week 45 | -47.27 (40.996) | -33.33 (50.319) | -25.91 (26.492) | -25.91 (38.680) | -61.59 (33.745) | -39.63 (39.211) | -47.19 (28.645) | -31.41 (39.716) | -27.07 (54.016)
  Week 46: number analyzed (Participants) | 12 | 32 | 10 | 27 | 12 | 31 | 7 | 29 | 11
  Week 46 | -42.11 (45.119) | -33.68 (49.356) | -34.27 (33.932) | -25.58 (38.019) | -58.81 (35.801) | -34.77 (38.757) | -49.76 (30.190) | -31.98 (39.640) | -28.89 (58.573)
  Week 47: number analyzed (Participants) | 12 | 32 | 9 | 27 | 12 | 31 | 7 | 30 | 13
  Week 47 | -40.77 (44.580) | -31.88 (48.778) | -25.60 (30.211) | -25.44 (39.798) | -59.01 (35.211) | -33.49 (39.386) | -48.45 (30.519) | -33.71 (38.282) | -25.86 (54.094)
  Week 48: number analyzed (Participants) | 12 | 32 | 9 | 27 | 12 | 30 | 7 | 29 | 13
  Week 48 | -36.53 (44.443) | -33.50 (48.912) | -30.33 (30.351) | -25.04 (38.230) | -61.01 (35.650) | -29.89 (38.681) | -51.75 (30.214) | -33.16 (40.239) | -29.29 (53.432)
  Week 49: number analyzed (Participants) | 12 | 31 | 10 | 27 | 12 | 30 | 7 | 30 | 12
  Week 49 | -36.35 (44.233) | -31.23 (48.493) | -34.64 (34.631) | -28.21 (41.352) | -61.21 (35.897) | -29.37 (38.374) | -48.17 (27.760) | -34.32 (41.018) | -29.80 (55.717)
  Week 50: number analyzed (Participants) | 12 | 31 | 10 | 27 | 12 | 29 | 7 | 30 | 12
  Week 50 | -36.14 (44.279) | -31.62 (50.758) | -32.01 (36.290) | -26.10 (40.637) | -59.59 (36.330) | -27.45 (38.441) | -50.18 (30.773) | -32.86 (40.330) | -31.15 (55.571)
  Week 51: number analyzed (Participants) | 12 | 30 | 10 | 27 | 11 | 29 | 7 | 30 | 12
  Week 51 | -34.31 (43.008) | -34.07 (51.575) | -30.83 (31.211) | -24.47 (39.779) | -60.72 (38.664) | -27.10 (39.790) | -48.66 (29.191) | -33.72 (40.790) | -30.75 (55.841)
  Week 52: number analyzed (Participants) | 12 | 30 | 9 | 27 | 12 | 29 | 7 | 30 | 12
  Week 52 | -35.06 (42.961) | -30.54 (49.791) | -33.29 (38.191) | -25.37 (39.165) | -61.83 (35.861) | -25.94 (43.683) | -50.89 (29.752) | -32.36 (40.612) | -30.50 (56.024)

46. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Weekly Average of Pruritus NRS (Numerical Rating Scale) ≥ 3 With a Baseline Pruritus NRS ≥ 3 From Baseline (Part 1)
Description: as for outcome 5
Time Frame: Baseline to weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, & 24
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 79 | 79
Percentage of participants
  Week 1 | 2.6 | 1.3 | 1.3 | 1.3 | 1.3
  Week 2 | 3.9 | 6.4 | 1.3 | 6.3 | 2.5
  Week 3 | 9.1 | 6.4 | 10.4 | 7.6 | 6.3
  Week 4 | 10.4 | 14.1 | 15.6 | 13.9 | 7.6
  Week 5 | 15.6 | 15.4 | 16.9 | 19.0 | 11.4
  Week 6 | 10.4 | 19.2 | 18.2 | 21.5 | 12.7
  Week 7 | 16.9 | 23.1 | 20.8 | 25.3 | 11.4
  Week 8 | 22.1 | 17.9 | 22.1 | 26.6 | 15.2
  Week 9 | 20.8 | 19.2 | 27.3 | 31.6 | 13.9
  Week 10 | 27.3 | 23.1 | 28.6 | 38.0 | 15.2
  Week 11 | 26.0 | 23.1 | 31.2 | 36.7 | 13.9
  Week 12 | 26.0 | 20.5 | 28.6 | 38.0 | 16.5
  Week 13 | 28.6 | 26.9 | 29.9 | 38.0 | 13.9
  Week 14 | 35.1 | 29.5 | 28.6 | 40.5 | 13.9
  Week 15 | 29.9 | 28.2 | 28.6 | 40.5 | 10.1
  Week 16 | 32.5 | 33.3 | 29.9 | 41.8 | 10.1
  Week 17 | 32.5 | 30.8 | 27.3 | 38.0 | 13.9
  Week 18 | 36.4 | 33.3 | 29.9 | 43.0 | 12.7
  Week 19 | 35.1 | 32.1 | 33.8 | 43.0 | 15.2
  Week 20 | 33.8 | 30.8 | 31.2 | 36.7 | 10.1
  Week 21 | 37.7 | 32.1 | 33.8 | 36.7 | 15.2
  Week 22 | 37.7 | 30.8 | 33.8 | 39.2 | 13.9
  Week 23 | 41.6 | 35.9 | 37.7 | 43.0 | 12.7
  Week 24 | 40.3 | 30.8 | 36.4 | 39.2 | 11.4

47. Secondary Outcome: Incidence Rate of Loss of EASI 50 (Part 2)
Description: The incidence rate of loss of EASI 50 is calculated for participants who achieved EASI 50 at re-randomization (week 24). The incidence rate is computed as the number of participants losing EASI 50 divided by total follow-up time. The follow-up time is defined as the duration from re-randomization (week 24) to either the first event date (loss of EASI 50) or censoring date for participants who had no events. The censoring date is defined as the earliest occurrence of: use of rescue medications and/or selected prohibited medications/ procedures impacting efficacy, or study discontinuation/ completion.
Time Frame: Week 24 to week 52
Population: Participants who reached EASI 50 at week 24 and re-randomized participants at week 24.
Measure: Number; unit: Events per patient-year
Arm/Group | 250 mg KY1005 Re-randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Events per patient-year | 0 | 0.272 | 0.188 | 0.089 | 0.165 | 0.071 | 0 | 0.193 | 0.145

48. Secondary Outcome: Incidence Rate of Loss of EASI 75 (Part 2)
Description: The incidence rate of loss of EASI 75 is calculated for participants who achieved EASI 75 at re-randomization (week 24). The incidence rate is computed as the number of participants losing EASI 75 divided by total follow-up time. The follow-up time is defined as the duration from re-randomization (week 24) to either the first event date (loss of EASI 75) or censoring date for participants who had no events. The censoring date is defined as the earliest occurrence of: use of rescue medications and/or selected prohibited medications/ procedures impacting efficacy, or study discontinuation/ completion.
Time Frame: Week 24 to week 52
Population: Participants who reached EASI 75 at week 24 and re-randomized participants at week 24.
Measure: Number; unit: Events per patient-year
Arm/Group | 250 mg KY1005 Re-randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 12 | 34 | 12 | 27 | 11 | 33 | 7 | 34 | 16
Events per patient-year | 0 | 0.587 | 0.375 | 0.486 | 0.395 | 0.446 | 0.351 | 0.573 | 0.646

49. Secondary Outcome: Incidence Rate of Loss of IGA 0/1 (Part 2)
Description: The incidence rate of loss of IGA 0/1 is calculated for participants who achieved IGA 0/1 at re-randomization (week 24). The incidence rate is computed as the number of participants losing IGA 0/1 divided by total follow-up time. The follow-up time is defined as the duration from re-randomization (week 24) to either the first event date (loss of IGA 0/1) or censoring date for participants who had no events. The censoring date is defined as the earliest occurrence of: use of rescue medications and/or selected prohibited medications/ procedures impacting efficacy, or study discontinuation/ completion.
Time Frame: Week 24 to week 68
Population: Participants who had IGA response 0 or 1 at week 24 and re-randomized at week 24.
Measure: Number; unit: Events per patient-year
Arm/Group | 250 mg KY1005 Re-randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 12 | 28 | 12 | 33 | 7 | 35 | 16
Events per patient-year | 1.267 | 1.039 | 0.981 | 1.930 | 1.154 | 1.045 | 1.096 | 1.790 | 0.244

50. Secondary Outcome: Serum KY1005 Concentration Assessed Throughout the Study (Part 1)
Time Frame: Baseline and at weeks 1, 2, 4, 8, 12, 16, 17, 20, & 24
Population: This analysis was conducted for Part 1 and includes participants who took at least one dose of KY1005. Only those participants with data available at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: (ug/ml)
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1)
Number analyzed (Participants) | 77 | 76 | 77 | 77
(ug/ml)
  Baseline: number analyzed (Participants) | 77 | 74 | 76 | 73
  Baseline | 0.00 (0.014) | 0.00 (0.014) | 0.01 (0.074) | 0.00 (0.000)
  Week 1: number analyzed (Participants) | 72 | 73 | 74 | 73
  Week 1 | 58.29 (24.674) | 30.49 (18.520) | 14.18 (5.060) | 8.49 (3.331)
  Week 2: number analyzed (Participants) | 65 | 69 | 67 | 70
  Week 2 | 47.56 (17.274) | 25.09 (9.041) | 13.56 (3.886) | 7.57 (2.947)
  Week 4: number analyzed (Participants) | 62 | 65 | 69 | 68
  Week 4 | 38.49 (22.532) | 19.00 (7.869) | 9.67 (3.728) | 5.09 (2.176)
  Week 8: number analyzed (Participants) | 53 | 48 | 56 | 61
  Week 8 | 37.67 (15.157) | 32.14 (16.502) | 15.07 (6.383) | 7.92 (3.263)
  Week 12: number analyzed (Participants) | 50 | 45 | 54 | 60
  Week 12 | 39.26 (33.847) | 34.67 (15.191) | 18.12 (8.439) | 9.22 (4.116)
  Week 16: number analyzed (Participants) | 49 | 48 | 49 | 52
  Week 16 | 40.12 (28.610) | 38.09 (13.536) | 18.39 (7.245) | 10.13 (4.515)
  Week 17: number analyzed (Participants) | 49 | 54 | 54 | 51
  Week 17 | 62.34 (28.081) | 64.64 (24.169) | 29.26 (11.659) | 16.79 (6.677)
  Week 20: number analyzed (Participants) | 49 | 49 | 54 | 56
  Week 20 | 37.92 (14.171) | 48.26 (30.691) | 19.31 (7.203) | 10.68 (3.715)
  Week 24: number analyzed (Participants) | 41 | 43 | 47 | 43
  Week 24 | 41.98 (23.087) | 43.81 (17.403) | 20.25 (10.575) | 11.07 (3.918)

51. Secondary Outcome: Serum KY1005 Concentration Assessed Throughout the Study (Part 2)
Time Frame: Baseline and at weeks 24, 25, 28, 32, 36, 40, 44, 48, & 52
Population: This analysis was conducted for Part 2 and includes participants who took at least one dose of KY1005. Only those participants with data available at specified timepoints are reported
Measure: Mean (Standard Deviation); unit: (ug/ml)
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2)
Number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 31 | 7 | 34
(ug/ml)
  Week 24: number analyzed (Participants) | 9 | 18 | 11 | 19 | 10 | 20 | 4 | 19
  Week 24 | 45.13 (15.842) | 36.68 (17.544) | 45.00 (14.568) | 43.17 (19.752) | 19.03 (9.612) | 19.48 (7.791) | 11.60 (1.383) | 11.10 (5.240)
  Week 25: number analyzed (Participants) | 12 | 28 | 10 | 23 | 10 | 24 | 4 | 24
  Week 25 | 73.54 (30.680) | 36.54 (20.508) | 71.25 (16.294) | 34.71 (14.551) | 31.07 (16.115) | 17.57 (7.504) | 15.90 (2.443) | 10.36 (5.145)
  Week 28: number analyzed (Participants) | 13 | 23 | 11 | 21 | 10 | 24 | 3 | 23
  Week 28 | 51.50 (25.454) | 17.59 (9.090) | 46.15 (15.782) | 25.22 (10.235) | 20.12 (11.820) | 10.03 (4.697) | 9.56 (3.485) | 6.66 (2.584)
  Week 32: number analyzed (Participants) | 11 | 20 | 10 | 15 | 9 | 18 | 3 | 21
  Week 32 | 44.41 (11.438) | 8.86 (5.074) | 41.50 (13.681) | 12.54 (5.943) | 20.99 (12.614) | 4.57 (2.463) | 9.40 (1.749) | 3.32 (1.588)
  Week 36: number analyzed (Participants) | 9 | 20 | 9 | 16 | 9 | 20 | 4 | 20
  Week 36 | 43.11 (18.965) | 5.41 (3.876) | 51.42 (18.946) | 7.80 (4.413) | 22.28 (18.101) | 2.85 (2.275) | 13.38 (2.128) | 1.77 (1.018)
  Week 40: number analyzed (Participants) | 9 | 20 | 9 | 18 | 8 | 23 | 5 | 20
  Week 40 | 45.19 (19.921) | 2.42 (1.660) | 43.79 (15.955) | 4.54 (2.929) | 19.09 (11.479) | 1.68 (1.669) | 10.95 (1.350) | 0.96 (0.748)
  Week 44: number analyzed (Participants) | 10 | 21 | 8 | 18 | 10 | 19 | 6 | 21
  Week 44 | 40.91 (12.068) | 1.04 (0.908) | 46.98 (24.015) | 2.62 (2.193) | 16.43 (7.302) | 0.82 (0.863) | 11.25 (2.607) | 0.57 (0.554)
  Week 48: number analyzed (Participants) | 11 | 18 | 8 | 19 | 9 | 19 | 6 | 20
  Week 48 | 41.43 (14.214) | 0.58 (0.507) | 43.63 (22.188) | 1.40 (1.727) | 17.80 (9.065) | 0.42 (0.483) | 11.12 (1.825) | 0.25 (0.305)
  Week 52: number analyzed (Participants) | 10 | 20 | 10 | 17 | 7 | 20 | 5 | 19
  Week 52 | 38.88 (11.526) | 0.56 (1.112) | 45.59 (22.447) | 0.55 (0.573) | 22.60 (8.225) | 0.19 (0.289) | 12.03 (3.775) | 0.11 (0.129)

52. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE) and Any Serious TEAE (Part 1)
Time Frame: Baseline through week 24
Population: Safety Analysis Part 1:Participants who took at least a dose of study treatment, including placebo up to Week 24. Analysis based on the SAF1 was based on the treatment received, regardless of assigned treatment according to the randomization
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 78 | 77 | 78 | 78
Percentage of participants
  Any Treatment Emergent Adverse Event | 66.2 | 66.7 | 67.5 | 67.9 | 60.3
  Any Serious Treatment Emergent Adverse Event | 2.6 | 0 | 1.3 | 6.4 | 1.3

53. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE) and Any Serious TEAE (Part 2)
Time Frame: Week 24 through week 68
Population: Safety Analysis Part 2: All re-randomized participants at Week 24 who took at least a dose of study treatment on/or after Week 24. Any analysis based on the SAF2 was based on the treatment at Week 24, regardless of treatment according to the randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg KY1005 Re-randomized From the 250mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2) Continued From Part 1 Placebo
Number analyzed (Participants) | 13 | 34 | 11 | 28 | 12 | 32 | 7 | 34 | 15
Percentage of participants
  Any Treatment Emergent Adverse Event | 84.6 | 67.6 | 63.6 | 78.6 | 66.7 | 87.5 | 57.1 | 67.6 | 66.7
  Any Serious Treatment Emergent Adverse Event | 7.7 | 2.9 | 0 | 7.1 | 8.3 | 0 | 0 | 0 | 0

54. Secondary Outcome: Percentage of Participants With Treatment-emergent ADA (Part 1)
Time Frame: Baseline through week 24
Population: The Full Analysis Set (FAS1) for Part 1 included all randomized participants up to Week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1)
Number analyzed (Participants) | 77 | 76 | 77 | 77
Percentage of participants | 2.6 | 6.4 | 13.2 | 32.1

55. Secondary Outcome: Percentage of Participants With Treatment-emergent ADA (Part 2)
Time Frame: Baseline through week 68
Population: The Full Analysis Set (FAS2) for Part 2 included all re-randomized at week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | 250 mg KY1005 Re-randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg Arm (Part 2) | 62.5 mg KY1005 Re-randomized From the 62.5 mg Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2)
Number analyzed (Participants) | 13 | 33 | 11 | 26 | 12 | 31 | 7 | 33
Percentage of participants | 7.7 | 9.1 | 9.1 | 19.2 | 0 | 35.5 | 28.6 | 42.4

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), all-cause mortality (deaths) were collected from the first dose of study treatment (Day 1) up to the last dose of the study treatment (Day 337)+ 140 days safety follow-up for each participant, up to 477 days
Description: Safety Analysis Part 1: Participants who received at least one dose of study treatment, including placebo, up to Week 24. Analysis based on SAF1 considered the treatment received, regardless of the assigned treatment according to randomization.
  Safety Analysis Part 2: All re-randomized participants at Week 24 who took at least one dose of study treatment on or after Week 24. Analysis based on SAF2 considered the treatment at Week 24, regardless of treatment according to the re-randomization.
Groups:
- Placebo (Part 2): Participants who completed Part 1 and who were responders (achieved ≥EASI 75 and/or who attained IGA 0/1 at Week 24 (Day 169) placebo received placebo Q4W from Week 24 to Week 52
Arm/Group | 250 mg (500 mg LD) KY1005 (Part 1) | 250 mg (no LD) KY1005 (Part 1) | 125 mg KY1005 (Part 1) | 62.5 mg KY1005 (Part 1) | Placebo (Part 1) | 250 mg KY1005 Re-Randomized From the 250 mg (LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) | Placebo (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78 | 0/77 | 0/78 | 0/78 | 0/13 | 0/34 | 0/11 | 0/28 | 0/12 | 0/32 | 0/7 | 0/34 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/77 | 0/78 | 1/77 | 5/78 | 1/78 | 1/13 | 1/34 | 0/11 | 2/28 | 1/12 | 0/32 | 0/7 | 0/34 | 0/15
Other Adverse Events (participants affected / at risk) | 42/77 | 39/78 | 39/77 | 41/78 | 41/78 | 11/13 | 21/34 | 7/11 | 19/28 | 8/12 | 27/32 | 4/7 | 21/34 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 250 mg (500 mg LD) KY1005 (Part 1) (N=77) | 250 mg (no LD) KY1005 (Part 1) (N=78) | 125 mg KY1005 (Part 1) (N=77) | 62.5 mg KY1005 (Part 1) (N=78) | Placebo (Part 1) (N=78) | 250 mg KY1005 Re-Randomized From the 250 mg (LD) Arm (Part 2) (N=13) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) (N=34) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) (N=11) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) (N=28) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) (N=12) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) (N=32) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) (N=7) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) (N=34) | Placebo (Part 2) (N=15)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | NA (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg (500 mg LD) KY1005 (Part 1) (N=77) | 250 mg (no LD) KY1005 (Part 1) (N=78) | 125 mg KY1005 (Part 1) (N=77) | 62.5 mg KY1005 (Part 1) (N=78) | Placebo (Part 1) (N=78) | 250 mg KY1005 Re-Randomized From the 250 mg (LD) Arm (Part 2) (N=13) | Placebo Re-Randomized From the 250 mg (LD) Arm (Part 2) (N=34) | 250 mg KY1005 Re-randomized From the 250 mg (No LD) Arm (Part 2) (N=11) | Placebo Re-Randomized From the 250 mg (No LD) Arm (Part 2) (N=28) | 125 mg KY1005 Re-randomized From the 125 mg Arm (Part 2) (N=12) | Placebo Re-randomized From the 125 mg KY1005 Arm (Part 2) (N=32) | 62.5 mg Re-Randomized From the 62.5 mg KY1005 Arm (Part 2) (N=7) | Placebo Re-randomized From the 62.5 mg Arm (Part 2) (N=34) | Placebo (Part 2) (N=15)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 7 (7) | 7 (7) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS INFECTED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 14 (19) | 6 (8) | 9 (12) | 5 (5) | 7 (10) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 5 (6) | 0 (0) | 3 (4) | 2 (3)
ORAL HERPES (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTITIS Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYURIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (3) | 4 (4) | 5 (6) | 5 (5) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 2 (3) | 4 (7) | 2 (3) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 4 (5) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIOSTITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 4 (4) | 4 (4) | 4 (4) | 7 (7) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TENSION HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 9 (10) | 16 (22) | 15 (19) | 13 (14) | 30 (43) | 6 (8) | 14 (21) | 3 (4) | 15 (19) | 1 (1) | 14 (17) | 1 (1) | 12 (13) | 4 (5)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT05131477/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT05131477/SAP_001.pdf